CLINICAL TRIAL: NCT05480800
Title: A Phase 1/2a, Observer-blind, Randomized, Controlled, Two-stage, Multi-country Study to Evaluate the Safety, Reactogenicity, and Immune Response of the Trivalent Vaccine Against Invasive Nontyphoidal Salmonella (iNTS) and Typhoid Fever in Healthy European and African Adults
Brief Title: A Study to Evaluate Safety, Reactogenicity, and Immune Response of GVGH iNTS-TCV Vaccine Against Invasive Nontyphoidal Salmonella and Typhoid Fever
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); Global Antimicrobial Resistance Innovation Fund-(GAMRIF) (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 216152; 2021-005178-25 (EudraCT Number)
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Salmonella Infections
MeSH Terms: conditions — Salmonella Infections | interventions — Meningococcal Vaccines; Boostrix; Vi polysaccharide vaccine, typhoid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Stage 1: Invasive nontyphoidal Salmonella (iNTS)-Typhoid conjugate vaccine (TCV) low dose group (Experimental): European participants were randomized to receive 3 doses of iNTS-TCV low dose vaccine and 3 doses of saline solution intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-typhoid conjugate vaccine (iNTS-TCV) low dose; Other: Saline
- Stage 1: iNTS-Generalized modules for membrane antigens (GMMA) + TCV low dose group (Active Comparator): European participants were randomized to receive 3 doses of iNTS-GMMA low dose vaccine and 3 doses of TCV low dose vaccine intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-generalized modules for membrane antigens vaccine (iNTS-GMMA) low dose; Biological: Typhoid conjugate vaccine (TCV) low dose
- Stage 1: iNTS-TCV full dose group (Experimental): European participants were randomized to receive 3 doses of iNTS-TCV full dose vaccine and 3 doses of saline solution intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-typhoid conjugate vaccine (iNTS-TCV) full dose; Other: Saline
- Stage 1: iNTS-GMMA + TCV full dose group (Active Comparator): European participants were randomized to receive 3 doses of iNTS-GMMA full dose vaccine and 3 doses of TCV full dose vaccine intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-generalized modules for membrane antigens vaccine (iNTS-GMMA) full dose; Biological: Typhoid conjugate vaccine (TCV) full dose
- Stage 1: Placebo group (Placebo Comparator): European participants were randomized to receive 3 doses of Placebo and 3 doses of saline solution intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Drug: Placebo; Other: Saline
- Stage 2: iNTS-TCV full dose group (Experimental): African participants were randomized to receive 3 doses of iNTS-TCV full dose vaccine and 3 doses of saline solution intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-typhoid conjugate vaccine (iNTS-TCV) full dose; Other: Saline
- Stage 2: iNTS-GMMA + TCV full dose group (Active Comparator): African participants were randomized to receive 3 doses of iNTS-GMMA full dose vaccine and 3 doses of TCV full dose intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
  Interventions: Biological: Invasive nontyphoidal Salmonella-generalized modules for membrane antigens vaccine (iNTS-GMMA) full dose; Biological: Typhoid conjugate vaccine (TCV) full dose
- Stage 2: Control group (Active Comparator): African participants were randomized to receive MENVEO as comparator and 1 dose of saline on Day 1, BOOSTRIX as comparator and 1 dose of saline on Day 57 and TYPHIM VI as comparator and 1 dose of saline on Day 169.
  Interventions: Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine; Combination Product: GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine; Combination Product: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine; Other: Saline

INTERVENTIONS:
Biological: Invasive nontyphoidal Salmonella-typhoid conjugate vaccine (iNTS-TCV) low dose — 3 doses of iNTS-TCV low dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-TCV low dose Group in Stage 1 (Europe).
  Arms: Stage 1: Invasive nontyphoidal Salmonella (iNTS)-Typhoid conjugate vaccine (TCV) low dose group
Biological: Invasive nontyphoidal Salmonella-generalized modules for membrane antigens vaccine (iNTS-GMMA) low dose — 3 doses of iNTS-GMMA low dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-GMMA and TCV low doses Group in Stage 1 (Europe).
  Arms: Stage 1: iNTS-Generalized modules for membrane antigens (GMMA) + TCV low dose group
Biological: Typhoid conjugate vaccine (TCV) low dose — 3 doses of TCV low dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-GMMA and TCV low doses Group in Stage 1 (Europe).
  Arms: Stage 1: iNTS-Generalized modules for membrane antigens (GMMA) + TCV low dose group
Biological: Invasive nontyphoidal Salmonella-typhoid conjugate vaccine (iNTS-TCV) full dose — 3 doses of iNTS-TCV full dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-TCV full dose Group in Stage 1 (Europe) and to participants in iNTS-TCV full dose Group in Stage 2 (Africa).
  Arms: Stage 1: iNTS-TCV full dose group; Stage 2: iNTS-TCV full dose group
Biological: Invasive nontyphoidal Salmonella-generalized modules for membrane antigens vaccine (iNTS-GMMA) full dose — 3 doses of iNTS-GMMA full dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-GMMA + TCV full dose Group in Stage 1 (Europe) and to participants in the iNTS-GMMA + TCV full dose Group in Stage 2 (Africa).
  Arms: Stage 1: iNTS-GMMA + TCV full dose group; Stage 2: iNTS-GMMA + TCV full dose group
Biological: Typhoid conjugate vaccine (TCV) full dose — 3 doses of TCV full dose vaccine administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the iNTS-GMMA + TCV full dose Group in Stage 1 (Europe) and to participants in the iNTS-GMMA + TCV full dose Group in Stage 2 (Africa).
  Arms: Stage 1: iNTS-GMMA + TCV full dose group; Stage 2: iNTS-GMMA + TCV full dose group
Biological: GSK's Meningococcal A, C, Y and W-135 conjugate vaccine — 1 dose of GSK's Meningococcal A, C, Y and W-135 conjugate vaccine administered intramuscularly at Day 1 to participants in the Control Group in Stage 2 (Africa).
  Other Names: MENVEO
  Arms: Stage 2: Control group
Combination Product: GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine — 1 dose of GSK's Tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine administered intramuscularly at Day 57 to participants in the Control Group in Stage 2 (Africa).
  Other Names: Boostrix
  Arms: Stage 2: Control group
Combination Product: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine — 1 dose of Sanofi Pasteur's Typhoid Vi polysaccharide vaccine administered intramuscularly at Day 169 to participants in the Control Group in Stage 2 (Africa).
  Other Names: TYPHIM Vi
  Arms: Stage 2: Control group
Drug: Placebo — 3 doses of Placebo administered intramuscularly at Day 1, Day 57, and Day 169 to participants in the Placebo Group in Stage 1 (Europe).
  Arms: Stage 1: Placebo group
Other: Saline — 3 doses of saline solution administered intramuscularly at Day 1, Day 57, and Day 169 to the participants.
  Arms: Stage 1: Invasive nontyphoidal Salmonella (iNTS)-Typhoid conjugate vaccine (TCV) low dose group; Stage 1: Placebo group; Stage 1: iNTS-TCV full dose group; Stage 2: Control group; Stage 2: iNTS-TCV full dose group

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity, and immune response induced by the GlaxoSmithKline Biologicals SA (GSK) Vaccines Institute for Global Health (GVGH) invasive nontyphoidal Salmonella-typhoid conjugate (iNTS-TCV) candidate vaccine to be administered for the first time in humans. The study intervention will be evaluated in European adults in Stage 1 (a 2-step staggered design) followed by African adults in Stage 2.

ELIGIBILITY:
Inclusion criteria

* Participants, who, in the opinion of the Investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history, clinical examination, and laboratory assessment.
* Participant satisfying screening requirements.
* A male or female between and including 18 and 50 years of age at the time of the first study intervention administration.
* Female participants of nonchildbearing potential may be enrolled in the study. Nonchildbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy, or post-menopause.
* Female participants of childbearing potential may be enrolled in the trial if the participant:
* Has practiced adequate contraception for 1 month prior to study intervention administration, and
* Has a negative pregnancy test on the day of study intervention administration, and
* Has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.
* Blood sample for simultaneous follicle-stimulating hormone (FSH) and estradiol levels may be collected at the discretion of the Investigator to confirm non-reproductive potential according to local laboratory reference range.
* Genetic testing for HLA-B27 will be performed at Screening and only participants with a negative result will be allowed to participate in the study*.

  * Only for Stage 1.
* For Malawi (Stage 2), the participant lives in Blantyre and has agreed to remain in Blantyre for the study duration.

Exclusion criteria Medical Conditions

* Known exposure to S. Typhi and nontyphoidal Salmonella confirmed by blood culture during the period starting 3 years prior to first study intervention administration confirmed using past medical history.
* History of any reaction or hypersensitivity associated with any component of the study interventions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Any clinically significant* hematological and/or biochemical laboratory abnormality.

  * The Investigator should use his/her clinical judgment to decide which abnormalities are clinically significant from the panel of tests in the list of safety assays.
* Clinical conditions representing a contraindication to IM injections and/or blood draws.
* Any behavioral or cognitive impairment or psychiatric disease that in the opinion of the Investigator, may interfere with the participant's ability to participate in the study.
* Confirmed positive COVID-19 polymerase chain reaction or lateral flow test during the period starting 28 days before the first administration of study vaccines (Day -28 to Day 1).
* Acute or chronic illness which may be severe enough to preclude participation.
* Any other clinical condition that, in the opinion of the Investigator, might pose additional risk to the participant due to participation in the study.
* All medical conditions will be assessed by the Investigator who may use his/her discretion to decide if the participant meets the exclusion criteria.

Prior/Concomitant Therapy

* History of receiving any typhoid vaccine (Ty21a, Vi capsular polysaccharide, or TCV) in the participant's life.
* History of receiving any investigational iNTS or GMMA vaccines in the participant's life.
* Use of any investigational or non-registered product other than the study interventions during the period beginning 30 days (Days -30 to 1) before the first dose of study interventions, or their planned use during the study period.
* A vaccine not foreseen by the study protocol administered during the period starting at 14 days before the first dose and ending 28 days after the last dose of study interventions administration*, with the exception of flu vaccines or COVID-19 vaccine.

  * In case emergency mass vaccination for an unforeseen public health threat (eg, a pandemic) is recommended and/or organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.

When regulations allow, the recommended time intervals for administration of these vaccines are at least 7 days before or 7 days after (at least 14 days before or 14 days after in case of live vaccines) each dose of study intervention administration.

* Administration of long-acting immune-modifying drugs at any time during the study period (eg, infliximab).
* Administration of Ig and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study interventions or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune modifying drugs during the period starting 3 months prior to the first study intervention dose(s). For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants. Inhaled and topical steroids are allowed.

Prior/Concurrent Clinical Study Experience

- Concurrently participating in another clinical trial, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (vaccine and drug).

Other Exclusions

* Pregnant or lactating female
* Female planning to become pregnant or planning to discontinue contraceptive precautions
* History of/current chronic alcohol consumption and/or drug abuse. This will be decided at the discretion of the Investigator. Chronic alcohol consumption is defined as one or more of the following:
* A prolonged period of frequent and heavy alcohol use
* The inability to control drinking once it has begun
* Physical dependence manifested by withdrawal symptoms when the individual stops using alcohol
* Tolerance or the need to use increasing amounts of alcohol to achieve the same effects
* A variety of social and/or legal problems arising from alcohol use.
* Any study personnel or their immediate dependents, family, or household members.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Edegem, Belgium
- GSK Investigational Site, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Started | 4 | 4 | 16 | 16 | 10 | 45 | 45 | 15
Completed | 4 | 4 | 14 | 15 | 10 | 45 | 43 | 15
Not Completed | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group | Total
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10 | 45 | 45 | 15 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.8 (2.5) | 35.8 (12.0) | 36.8 (11.1) | 33.1 (11.3) | 34.7 (9.5) | 28.2 (6.3) | 28.5 (6.3) | 29.7 (9.1) | 30.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 11 | 10 | 10 | 26 | 23 | 5 | 90
  Male | 0 | 3 | 5 | 6 | 0 | 19 | 22 | 10 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 15 | 16 | 9 | 0 | 0 | 0 | 48
  Black or African American | 0 | 0 | 0 | 0 | 0 | 45 | 45 | 14 | 104
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Stage 1 and Stage 2: Number of Participants With Any SAEs
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement. Any = occurrence of the event regardless of intensity grade.
Time Frame: From 28 days after the third study intervention administration (Day 197) up to study end (Day 337)
Population: The analysis was performed on the exposed set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10 | 45 | 45 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

2. Secondary Outcome: Stage 1 and Stage 2: Number of Participants With Any AEs/SAEs Leading to Withdrawal From the Study
Description: Any AEs including SAEs that lead to withdrawal from the study are considered under this outcome measure. A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact. Any = occurrence of the event regardless of intensity grade.
Time Frame: From 28 days after the third study intervention administration (Day 197) up to study end (Day 337)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10 | 45 | 45 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Stage 1: Geometric Mean Concentrations (GMCs) of Anti-serotype Specific Immunoglobulin G (IgG) in Participants and Between Group Ratios for Anti-Vi Antigen (Ag) Total IgG
Description: Anti-Vi antigen (Ag) total IgG GMCs were assessed. Blood samples were collected at specified timepoint for each component as measured by Enzyme-Linked Immunosorbent Assay (ELISA). The lower limit of quantification (LLOQ) for antibody concentrations was >=2.2 microgram per milliliter (µg/mL). In case the measured antibody concentration fell below 2.2 µg/mL, a value of half the LLOQ value was imputed.
Time Frame: At Days 1, 57, and 169 (before each study intervention administration) and at Days 29, 85, and 197 (28 days after each study intervention administration)
Population: The analysis was performed on the Per Protocol Set (PPS), that included all eligible participants who received all doses as per protocol, had immunogenicity results post-dose, complied with dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
microgram per milliliter (µg/mL)
  Anti-Vi Ag total IgG, Day 1: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-Vi Ag total IgG, Day 1 | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ (lower limit of quantification). | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ. | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ. | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ. | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ.
  Anti-Vi Ag total IgG, Day 29: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-Vi Ag total IgG, Day 29 | 30.29 [13.50 to 67.95] | 68.87 [1.73 to 2741.00] | 43.55 [18.51 to 102.49] | 66.48 [37.31 to 118.46] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs for this group as all participants were below LLOQ.
  Anti-Vi Ag total IgG, Day 57: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-Vi Ag total IgG, Day 57 | 23.28 [16.49 to 32.89] | 53.95 [2.37 to 1226.99] | 25.99 [9.86 to 68.50] | 51.01 [27.55 to 94.46] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs for this group as all participants were below LLOQ.
  Anti-Vi Ag total IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-Vi Ag total IgG, Day 85 | 30.52 [14.75 to 63.13] | 51.71 [3.42 to 781.48] | 34.02 [16.67 to 69.44] | 51.65 [31.18 to 85.55] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs for this group as all participants were below LLOQ.
  Anti-Vi Ag total IgG, Day 169: number analyzed (Participants) | 4 | 2 | 13 | 14 | 10
  Anti-Vi Ag total IgG, Day 169 | 13.61 [4.28 to 43.23] | 14.11 [0.22 to 10265.73] | 15.76 [8.14 to 30.48] | 20.69 [12.68 to 33.76] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs for this group as all participants were below LLOQ.
  Anti-Vi Ag total IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-Vi Ag total IgG, Day 197 | 20.19 [1.48 to 275.08] | 17.43 [0.01 to 26224.47] | 31.84 [16.24 to 62.43] | 35.24 [23.65 to 52.49] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs for this group as all participants were below LLOQ.
Statistical Analysis 1: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-Vi Ag IgG, Day 29; Test type: Other — The statistical analyses performed for the study objectives were descriptive. No success criteria were defined for the statistical analyses conducted in this study; ANOVA; Unadjusted GMR = 0.44, 95% CI [0.06 to 3.43] — The Unadjusted Geometric Mean Ratio (GMR) is the ratio of the geometric means of two groups being compared. Results were based on a linear model for a visit with fixed effect for treatment
Statistical Analysis 2: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG, Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.66, 95% CI [0.25 to 1.70] — The Unadjusted GMR is the ratio of the geometric means of two groups being compared. Results were based on a linear model for a visit with fixed effect for treatment
Statistical Analysis 3: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-Vi Ag IgG, Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.43, 95% CI [0.06 to 2.94] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG, Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.51, 95% CI [0.19 to 1.37] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-Vi Ag IgG, Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.59, 95% CI [0.13 to 2.65] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG, Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.66, 95% CI [0.30 to 1.43] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-Vi Ag IgG, Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.96, 95% CI [0.18 to 5.12] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG, Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.76, 95% CI [0.36 to 1.60] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-Vi Ag IgG, Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.16, 95% CI [0.23 to 5.79] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG, Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.90, 95% CI [0.44 to 1.84] — [estimate comment as in outcome 3, analysis 2]

4. Secondary Outcome: Stage 1: GMCs of Anti-serotype Specific IgG in Participants and Between Group Ratios for Anti-S. Typhimurium OAg Total IgG and Anti-S. Enteritidis OAg Total IgG
Description: Anti-S. Typhimurium OAg total IgG, Anti-S. Enteritidis OAg total IgG GMCs were assessed. Blood samples were collected at specified timepoint for each component as measured by Enzyme-Linked Immunosorbent Assay (ELISA).
Time Frame: as for outcome 3
Population: The analysis was performed on the PPS. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter (EU/mL)
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
ELISA units per milliliter (EU/mL)
  Anti-S.Typhimurium OAg IgG, Day 1: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-S.Typhimurium OAg IgG, Day 1 | 20.25 [3.23 to 126.95] | 49.45 [0.68 to 3599.82] | 94.10 [34.63 to 255.69] | 124.02 [54.83 to 280.53] | 52.23 [19.31 to 141.31]
  Anti-S.Typhimurium OAg IgG, Day 29: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-S.Typhimurium OAg IgG, Day 29 | 494.50 [80.16 to 3050.49] | 169.25 [4.35 to 6586.95] | 1426.07 [777.69 to 2615.03] | 1505.55 [815.65 to 2778.99] | 52.86 [19.93 to 140.20]
  Anti-S.Typhimurium OAg IgG, Day 57: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Typhimurium OAg IgG, Day 57 | 423.33 [81.46 to 2200.08] | 139.78 [5.42 to 3604.75] | 1075.57 [466.12 to 2481.85] | 1203.79 [589.73 to 2457.26] | 58.38 [16.45 to 207.16]
  Anti-S.Typhimurium OAg IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Typhimurium OAg IgG, Day 85 | 410.29 [87.67 to 1920.18] | 243.42 [3.18 to 18606.83] | 1129.27 [497.20 to 2564.86] | 1478.01 [804.57 to 2715.11] | 68.07 [17.22 to 269.09]
  Anti-S.Typhimurium OAg IgG, Day 169: number analyzed (Participants) | 4 | 2 | 13 | 14 | 10
  Anti-S.Typhimurium OAg IgG, Day 169 | 272.19 [43.10 to 1718.88] | 109.20 [0.00 to 1040000000000] | 703.74 [296.98 to 1667.63] | 951.71 [498.59 to 1816.63] | 75.80 [21.92 to 262.14]
  Anti-S.Typhimurium OAg IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-S.Typhimurium OAg IgG, Day 197 | 249.07 [21.83 to 2842.34] | 163.07 [0.00 to 1190000000000] | 1005.05 [445.54 to 2267.20] | 1176.88 [719.47 to 1925.10] | 73.43 [21.98 to 245.25]
  Anti-S.Enteritidis OAg IgG, Day 1: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-S.Enteritidis OAg IgG, Day 1 | 67.85 [6.04 to 761.69] | 42.77 [0.32 to 5784.66] | 125.64 [47.39 to 333.09] | 115.74 [46.32 to 289.22] | 57.08 [21.97 to 148.25]
  Anti-S.Enteritidis OAg IgG, Day 29: number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
  Anti-S.Enteritidis OAg IgG, Day 29 | 920.64 [104.11 to 8141.15] | 169.46 [0.32 to 90734.61] | 1648.46 [1023.81 to 2654.22] | 1387.16 [587.94 to 3272.77] | 56.62 [21.49 to 149.13]
  Anti-S.Enteritidis OAg IgG, Day 57: number analyzed (Participants) | 4 | 3 | 12 | 16 | 9
  Anti-S.Enteritidis OAg IgG, Day 57 | 832.83 [110.24 to 6291.99] | 141.59 [0.42 to 47560.41] | 1454.26 [801.81 to 2637.64] | 1076.32 [400.41 to 2893.21] | 65.49 [18.13 to 236.58]
  Anti-S.Enteritidis OAg IgG, Day 85: number analyzed (Participants) | 4 | 4 | 12 | 16 | 9
  Anti-S.Enteritidis OAg IgG, Day 85 | 882.68 [132.51 to 5879.62] | 209.03 [0.88 to 49901.51] | 1436.56 [779.81 to 2646.42] | 1267.65 [511.67 to 3140.56] | 79.79 [18.55 to 343.09]
  Anti-S.Enteritidis OAg IgG, Day 169: number analyzed (Participants) | 4 | 4 | 13 | 16 | 10
  Anti-S.Enteritidis OAg IgG, Day 169 | 557.81 [78.28 to 3975.01] | 42.14 [0.01 to 162000] | 903.37 [487.13 to 1675.30] | 729.86 [255.41 to 2085.64] | 75.96 [20.72 to 278.48]
  Anti-S.Enteritidis OAg IgG, Day 197 | 451.36 [22.54 to 9036.65] | 81.17 [0.87 to 7578.12] | 1168.56 [642.31 to 2125.99] | 855.62 [356.65 to 2052.67] | 73.74 [20.17 to 269.56]
Statistical Analysis 1: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Typhimurium OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 2.92, 95% CI [0.48 to 17.80] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.95, 95% CI [0.41 to 2.19] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Typhimurium OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 3.03, 95% CI [0.43 to 21.45] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.89, 95% CI [0.33 to 2.45] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Typhimurium OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.69, 95% CI [0.26 to 10.96] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.76, 95% CI [0.29 to 2.00] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Typhimurium OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 2.49, 95% CI [0.24 to 26.30] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.74, 95% CI [0.26 to 2.11] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Typhimurium OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.53, 95% CI [0.19 to 12.41] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.85, 95% CI [0.34 to 2.15] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 11: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Enteritidis OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 5.43, 95% CI [0.61 to 48.17] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 12: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.19, 95% CI [0.43 to 3.26] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 13: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Enteritidis OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 5.88, 95% CI [0.58 to 59.45] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 14: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.35, 95% CI [0.41 to 4.45] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 15: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Enteritidis OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 4.22, 95% CI [0.48 to 37.19] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 16: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.13, 95% CI [0.37 to 3.48] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 17: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Enteritidis OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 13.24, 95% CI [1.02 to 172.55] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 18: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.24, 95% CI [0.40 to 3.88] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 19: Comparison: Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group vs Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group; Anti-S.Enteritidis OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 5.56, 95% CI [0.53 to 58.61] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 20: Comparison: Stage 1: iNTS-TCV Full Dose Group vs Stage 1: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.37, 95% CI [0.48 to 3.86] — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Stage 1: Geometric Mean Ratios (GMRs) for Anti-serotype Specific Immunoglobulin G (IgG) Concentrations
Description: Anti-Vi antigen (Ag) total IgG, Anti-S. Typhimurium OAg total IgG, Anti-S. Enteritidis OAg total IgG within-participant GMRs were assessed. Blood samples were collected at specified timepoint for each component as measured by ELISA. Within participant GMRs were calculated as ratio of concentration in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At 28 days after each study intervention administration compared to each study intervention administration baseline (Day 29 versus Day 1, Day 85 versus Day 57 and Day 197 versus Day 169)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
Ratio
  Anti-Vi Ag total IgG, Day 29 | 27.53 [12.27 to 61.77] | 62.61 [1.57 to 2491.81] | 39.60 [16.83 to 93.18] | 60.44 [33.92 to 107.69] | 1.00 [1.00 to 1.00]
  Anti-Vi Ag total IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-Vi Ag total IgG, Day 85 | 1.31 [0.80 to 2.14] | 0.96 [0.47 to 1.96] | 1.31 [0.87 to 1.97] | 1.01 [0.78 to 1.31] | 1.00 [1.00 to 1.00]
  Anti-Vi Ag total IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-Vi Ag total IgG, Day 197 | 1.96 [0.49 to 7.78] | 1.24 [0.60 to 2.55] | 1.99 [1.38 to 2.89] | 1.70 [1.38 to 2.10] | 1.00 [1.00 to 1.00]
  Anti-S.Typhimurium OAg IgG. Day 29 | 24.42 [11.30 to 52.75] | 3.42 [0.48 to 24.20] | 15.15 [5.57 to 41.26] | 12.14 [6.83 to 21.58] | 1.01 [0.94 to 1.09]
  Anti-S.Typhimurium OAg IgG. Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Typhimurium OAg IgG. Day 85 | 0.97 [0.63 to 1.50] | 1.74 [0.44 to 6.87] | 1.05 [0.86 to 1.28] | 1.23 [0.89 to 1.69] | 1.17 [0.97 to 1.40]
  Anti-S.Typhimurium OAg IgG. Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-S.Typhimurium OAg IgG. Day 197 | 1.47 [0.80 to 2.71] | 1.49 [1.14 to 1.95] | 1.20 [1.01 to 1.44] | 1.24 [0.93 to 1.65] | 0.97 [0.90 to 1.04]
  Anti-S.Enteritidis OAg IgG Day 29 | 13.57 [3.76 to 48.93] | 3.96 [0.67 to 23.52] | 13.12 [5.41 to 31.80] | 11.98 [6.57 to 21.86] | 0.99 [0.93 to 1.06]
  Anti-S.Enteritidis OAg IgG Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Enteritidis OAg IgG Day 85 | 1.06 [0.90 to 1.24] | 1.48 [0.59 to 3.67] | 0.99 [0.86 to 1.14] | 1.18 [0.82 to 1.69] | 1.22 [0.97 to 1.53]
  Anti-S.Enteritidis OAg IgG Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-S.Enteritidis OAg IgG Day 197 | 1.29 [0.68 to 2.45] | 1.93 [0.05 to 79.54] | 1.15 [1.03 to 1.28] | 1.17 [0.92 to 1.49] | 0.97 [0.95 to 0.99]

6. Secondary Outcome: Stage 1: Number of Participants Achieving at Least a 4 Fold Rise in Anti Serotype Specific Immunoglobulin G (IgG) Antibody Concentration for Each Antigen (Ag)
Description: Anti-Vi Ag total IgG, Anti-S. Typhimurium OAg total IgG, Anti-S. Enteritidis OAg total IgG antibody concentrations were assessed. Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: At Days 29, 85, and 197 (28 days after each study intervention administration) compared to Day 1 (first study intervention administration)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
Participants
  Anti-Vi Ag IgG, Day 29 | 4 | 3 | 13 | 16 | 0
  Anti-Vi Ag IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-Vi Ag IgG, Day 85 | 4 | 3 | 10 | 14 | 0
  Anti-Vi Ag IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-Vi Ag IgG, Day 197 | 2 | 2 | 10 | 14 | 0
  Anti-S.Typhimurium OAg IgG, Day 29 | 4 | 1 | 13 | 15 | 0
  Anti-S.Typhimurium OAg IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Typhimurium OAg IgG, Day 85 | 4 | 2 | 8 | 14 | 1
  Anti-S.Typhimurium OAg IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-S.Typhimurium OAg IgG, Day 197 | 3 | 1 | 6 | 10 | 1
  Anti-S.Enteritidis OAg IgG, Day 29 | 4 | 1 | 11 | 12 | 0
  Anti-S.Enteritidis OAg IgG, Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Anti-S.Enteritidis OAg IgG, Day 85 | 4 | 2 | 7 | 11 | 1
  Anti-S.Enteritidis OAg IgG, Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Anti-S.Enteritidis OAg IgG, Day 197 | 3 | 1 | 4 | 10 | 1

7. Secondary Outcome: Stage 1: Number of Participants With Anti-Vi Ag IgG Antibody Concentrations Greater Than or Equal to (>=) 4.3 Micrograms Per Milliliter (µg/mL)
Description: Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: At Days 1, 57 and 169 (before each study intervention administration) and at Days 29, 85 and 197 (28 days after each study intervention administration)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 16 | 16 | 10
Participants
  Day 1 (pre-Dose 1) | 0 | 0 | 0 | 0 | 0
  Day 29 | 4 | 3 | 14 | 16 | 0
  Day 57 (pre-Dose 2): number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Day 57 (pre-Dose 2) | 4 | 3 | 9 | 14 | 0
  Day 85: number analyzed (Participants) | 4 | 3 | 12 | 14 | 9
  Day 85 | 4 | 3 | 12 | 14 | 0
  Day 169 (pre-Dose 3): number analyzed (Participants) | 4 | 2 | 13 | 14 | 10
  Day 169 (pre-Dose 3) | 4 | 2 | 11 | 14 | 0
  Day 197: number analyzed (Participants) | 3 | 2 | 11 | 14 | 10
  Day 197 | 3 | 2 | 11 | 14 | 0

8. Secondary Outcome: Stage 2: GMCs of Anti-serotype Specific IgG in Participants and Between Group Ratios for Anti-Vi Ag Total IgG
Description: Anti-Vi Ag total IgG GMCs and between group ratios were assessed. Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Stage 2: iNTS-GMMA + TCV Full Dose Group: African participants were randomized to receive 3 doses of iNTS-GMMA full dose vaccineand 3 doses of TCV full dose intramuscularly, in different arms, on Day 1, Day 57 and Day 169.
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 44 | 15
µg/mL
  Anti-Vi Ag total IgG, Day 1 | 1.43 [1.20 to 1.70] | 1.38 [1.13 to 1.69] | 1.56 [1.11 to 2.19]
  Anti-Vi Ag total IgG, Day 29 | 148.98 [103.31 to 214.83] | 161.68 [107.38 to 243.46] | 1.55 [1.04 to 2.33]
  Anti-Vi Ag total IgG, Day 57 | 96.93 [67.00 to 140.23] | 104.38 [69.77 to 156.16] | 1.60 [1.01 to 2.53]
  Anti-Vi Ag total IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-Vi Ag total IgG, Day 85 | 96.94 [72.03 to 130.48] | 101.92 [72.02 to 144.24] | 1.65 [1.08 to 2.52]
  Anti-Vi Ag total IgG, Day 169: number analyzed (Participants) | 41 | 38 | 14
  Anti-Vi Ag total IgG, Day 169 | 41.83 [29.43 to 59.46] | 53.65 [34.97 to 82.32] | 1.88 [1.18 to 2.99]
  Anti-Vi Ag total IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-Vi Ag total IgG, Day 197 | 65.43 [51.01 to 83.92] | 69.82 [50.09 to 97.30] | 18.60 [8.28 to 41.76]
Statistical Analysis 1: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.92, 95% CI [0.54 to 1.58] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 2: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.93, 95% CI [0.54 to 1.59] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.95, 95% CI [0.61 to 1.49] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.78, 95% CI [0.45 to 1.34] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-Vi Ag IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.94, 95% CI [0.63 to 1.40] — [estimate comment as in outcome 3, analysis 2]

9. Secondary Outcome: Stage 2: GMCs of Anti-serotype Specific IgG in Participants and Between Group Ratios for Anti-S. Typhimurium OAg Total IgG and Anti-S. Enteritidis OAg Total IgG
Description: Anti-S. Typhimurium OAg total IgG and Anti-S. Enteritidis OAg total IgG GMCs and between group ratios were assessed. Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 44 | 15
EU/mL
  Anti-S.Typhimurium OAg IgG, Day 1 | 246.02 [167.63 to 361.07] | 490.94 [378.78 to 636.31] | 392.99 [273.90 to 563.87]
  Anti-S.Typhimurium OAg IgG, Day 29 | 1591.68 [1117.07 to 2267.94] | 2585.81 [2024.74 to 3302.35] | 446.22 [290.49 to 685.45]
  Anti-S.Typhimurium OAg IgG, Day 57 | 1159.50 [806.72 to 1666.56] | 1794.69 [1419.63 to 2268.85] | 483.46 [329.52 to 709.32]
  Anti-S.Typhimurium OAg IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Typhimurium OAg IgG, Day 85 | 1102.67 [771.64 to 1575.70] | 1765.79 [1395.81 to 2233.85] | 545.05 [355.58 to 835.46]
  Anti-S.Typhimurium OAg IgG, Day 169: number analyzed (Participants) | 41 | 38 | 14
  Anti-S.Typhimurium OAg IgG, Day 169 | 870.80 [552.07 to 1373.57] | 1248.95 [979.10 to 1593.18] | 565.73 [349.09 to 916.82]
  Anti-S.Typhimurium OAg IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Typhimurium OAg IgG, Day 197 | 992.82 [645.92 to 1526.03] | 1748.80 [1359.79 to 2249.09] | 542.87 [340.01 to 866.75]
  Anti-S.Enteritidis OAg IgG, Day 1 | 363.08 [228.49 to 576.96] | 376.17 [270.58 to 522.95] | 394.19 [193.54 to 802.88]
  Anti-S.Enteritidis OAg IgG, Day 29 | 1884.94 [1272.38 to 2792.41] | 2295.38 [1642.33 to 3208.10] | 457.08 [209.54 to 997.03]
  Anti-S.Enteritidis OAg IgG, Day 57 | 1527.50 [1030.99 to 2263.13] | 1581.75 [1153.18 to 2169.60] | 470.88 [214.12 to 1035.51]
  Anti-S.Enteritidis OAg IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Enteritidis OAg IgG, Day 85 | 1604.28 [1109.24 to 2320.23] | 1555.91 [1134.43 to 2133.97] | 456.04 [215.01 to 967.26]
  Anti-S.Enteritidis OAg IgG, Day 169: number analyzed (Participants) | 41 | 38 | 14
  Anti-S.Enteritidis OAg IgG, Day 169 | 946.93 [646.79 to 1386.34] | 1015.74 [727.61 to 1417.95] | 408.69 [190.40 to 877.23]
  Anti-S.Enteritidis OAg IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Enteritidis OAg IgG, Day 197 | 1093.84 [757.63 to 1579.27] | 1327.68 [972.03 to 1813.45] | 423.08 [213.16 to 839.75]
Statistical Analysis 1: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Adjusted GMR = 0.95, 95% CI [0.69 to 1.32] — Results based on a linear mixed model with fixed effects; denominator degrees of freedom adjusted using Satterthwaite's method; Heterogeneity was observed at baseline for S. Typhimurium in Africa between iNTS - GMMA + TCV Full dose and iNTS-TCV Ful dose, which influenced other timepoints. Hence, adjusted GMRs are presented
Statistical Analysis 2: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Adjusted GMR = 1.01, 95% CI [0.74 to 1.37] — [estimate comment as in outcome 9, analysis 1]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Adjusted GMR = 1.04, 95% CI [0.77 to 1.41] — [estimate comment as in outcome 9, analysis 1]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Adjusted GMR = 1.20, 95% CI [0.81 to 1.77] — [estimate comment as in outcome 9, analysis 1]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Typhimurium OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; Mixed Models Analysis; Adjusted GMR = 0.97, 95% CI [0.65 to 1.44] — [estimate comment as in outcome 9, analysis 1]; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 29; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.82, 95% CI [0.49 to 1.37] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 7: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 57; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.97, 95% CI [0.59 to 1.59] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 8: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 85; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 1.03, 95% CI [0.64 to 1.67] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 9: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 169; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.93, 95% CI [0.56 to 1.54] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 10: Comparison: Stage 2: iNTS-TCV Full Dose Group vs Stage 2: iNTS-GMMA + TCV Full Dose Group; Anti-S.Enteritidis OAg IgG Day 197; Test type: Other — [test comment as in outcome 3, analysis 1]; ANOVA; Unadjusted GMR = 0.82, 95% CI [0.51 to 1.33] — [estimate comment as in outcome 3, analysis 2]

10. Secondary Outcome: Stage 2: GMRs for Anti-serotype Specific Immunoglobulin G (IgG) Concentrations
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 44 | 15
Ratio
  Anti-Vi Ag total IgG, Day 29 | 104.51 [77.39 to 141.12] | 116.84 [79.82 to 171.01] | 1.00 [0.74 to 1.34]
  Anti-Vi Ag total IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-Vi Ag total IgG, Day 85 | 1.05 [0.92 to 1.20] | 0.91 [0.83 to 1.00] | 1.03 [0.92 to 1.16]
  Anti-Vi Ag total IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-Vi Ag total IgG, Day 197 | 1.56 [1.30 to 1.88] | 1.37 [1.10 to 1.69] | 9.89 [5.14 to 19.04]
  Anti-S.Typhimurium OAg IgG. Day 29 | 6.47 [4.97 to 8.42] | 5.27 [4.12 to 6.73] | 1.14 [0.83 to 1.55]
  Anti-S.Typhimurium OAg IgG. Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Typhimurium OAg IgG. Day 85 | 1.00 [0.92 to 1.10] | 0.97 [0.89 to 1.06] | 1.13 [0.89 to 1.42]
  Anti-S.Typhimurium OAg IgG. Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Typhimurium OAg IgG. Day 197 | 1.14 [1.04 to 1.25] | 1.41 [1.18 to 1.70] | 0.96 [0.81 to 1.14]
  Anti-S.Enteritidis OAg IgG Day 29 | 5.19 [3.44 to 7.83] | 6.10 [4.47 to 8.33] | 1.16 [0.82 to 1.65]
  Anti-S.Enteritidis OAg IgG Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Enteritidis OAg IgG Day 85 | 1.04 [0.94 to 1.15] | 0.99 [0.90 to 1.10] | 0.97 [0.83 to 1.13]
  Anti-S.Enteritidis OAg IgG Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Enteritidis OAg IgG Day 197 | 1.16 [1.00 to 1.34] | 1.34 [1.11 to 1.62] | 1.04 [0.86 to 1.25]

11. Secondary Outcome: Stage 2: Number of Participants Achieving at Least a 4 Fold Rise in Anti Serotype Specific Immunoglobulin G (IgG) Antibody Concentration for Each Antigen (Ag)
Description: as for outcome 6
Time Frame: At Days 29, 85, and 197 (28 days after each study intervention administration) compared to Day 1 (first study intervention administration baseline)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 44 | 15
Participants
  Anti-Vi Ag IgG, Day 29 | 44 | 43 | 0
  Anti-Vi Ag IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-Vi Ag IgG, Day 85 | 44 | 42 | 1
  Anti-Vi Ag IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-Vi Ag IgG, Day 197 | 41 | 37 | 9
  Anti-S.Typhimurium OAg IgG, Day 29 | 33 | 27 | 1
  Anti-S.Typhimurium OAg IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Typhimurium OAg IgG, Day 85 | 22 | 16 | 1
  Anti-S.Typhimurium OAg IgG, 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Typhimurium OAg IgG, 197 | 23 | 16 | 1
  Anti-S.Enteritidis OAg IgG, 29 | 23 | 27 | 1
  Anti-S.Enteritidis OAg IgG, Day 85: number analyzed (Participants) | 44 | 43 | 15
  Anti-S.Enteritidis OAg IgG, Day 85 | 21 | 18 | 2
  Anti-S.Enteritidis OAg IgG, Day 197: number analyzed (Participants) | 41 | 37 | 14
  Anti-S.Enteritidis OAg IgG, Day 197 | 17 | 16 | 0

12. Secondary Outcome: Stage 2: Number of Participants With Anti-Vi Ag IgG Antibody Concentrations >= 4.3 µg/mL
Description: Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: as for outcome 7
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 44 | 15
Participants
  Day 1 | 4 | 3 | 3
  Day 29 | 45 | 44 | 3
  Day 57 | 45 | 44 | 3
  Day 85: number analyzed (Participants) | 44 | 43 | 15
  Day 85 | 44 | 43 | 3
  Day 169: number analyzed (Participants) | 41 | 38 | 14
  Day 169 | 41 | 37 | 3
  Day 197: number analyzed (Participants) | 41 | 37 | 14
  Day 197 | 41 | 37 | 12

13. Primary Outcome: Stage 1: Number of Participants With Any Solicited Administration Site Events After the First Study Intervention Administration
Description: The solicited administration site events included redness (erythema), pain, and swelling. Data for solicited administration site events is presented for each intervention administered in each arm group. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-first vaccination on Day 1)
Population: The analysis was performed on the Solicited safety set, which included all participants who received first dose of the study intervention and who had solicited safety data in the 7 days following first intervention. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants
  Redness, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV low dose | 1 | 0 | 0 | 0 | 0
  Redness, Saline: number analyzed (Participants) | 4 | 0 | 16 | 0 | 10
  Redness, Saline | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose | 0 | 0 | 0 | 0 | 0
  Redness, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Redness, TCV low dose | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 16 | 0 | 0
  Redness, iNTS-TCV full dose | 0 | 0 | 4 | 0 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Redness, iNTS-GMMA full dose | 0 | 0 | 0 | 5 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Redness, TCV full dose | 0 | 0 | 0 | 0 | 0
  Redness, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Redness, Placebo | 0 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose | 4 | 0 | 0 | 0 | 0
  Pain, saline: number analyzed (Participants) | 4 | 0 | 16 | 0 | 10
  Pain, saline | 0 | 0 | 1 | 0 | 3
  Pain, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Pain, iNTS-GMMA low dose | 0 | 4 | 0 | 0 | 0
  Pain, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Pain, TCV low dose | 0 | 1 | 0 | 0 | 0
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 16 | 0 | 0
  Pain, iNTS-TCV full dose | 0 | 0 | 16 | 0 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Pain, iNTS-GMMA full dose | 0 | 0 | 0 | 16 | 0
  Pain, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Pain, TCV full dose | 0 | 0 | 0 | 1 | 0
  Pain, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Pain, Placebo | 0 | 0 | 0 | 0 | 3
  Swelling, iNTS-TCV Low: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Swelling, iNTS-TCV Low | 1 | 0 | 0 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 4 | 0 | 16 | 0 | 10
  Swelling, saline | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose | 0 | 1 | 0 | 0 | 0
  Swelling, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Swelling, TCV low dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 16 | 0 | 0
  Swelling, iNTS-TCV full dose | 0 | 0 | 4 | 0 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Swelling, iNTS-GMMA full dose | 0 | 0 | 0 | 3 | 0
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 16 | 0
  Swelling, TCV full dose | 0 | 0 | 0 | 0 | 0
  Swelling, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Swelling, Placebo | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Stage 1: Number of Participants With Any Solicited Administration Site Events After the Second Study Intervention Administration
Description: The solicited administration site events included redness (Erythema), pain and swelling. Data for solicited administration site events is presented for each intervention administered in each arm group. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-second vaccination on Day 57)
Population: The analysis was performed on the Solicited safety set, which included all participants who received second dose of the study intervention and who had solicited safety data in the 7 days following second intervention. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 15 | 15 | 10
Participants
  Redness, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV low dose | 0 | 0 | 0 | 0 | 0
  Redness, Saline: number analyzed (Participants) | 4 | 0 | 15 | 0 | 10
  Redness, Saline | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose | 0 | 0 | 0 | 0 | 0
  Redness, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Redness, TCV low dose | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 15 | 0 | 0
  Redness, iNTS-TCV full dose | 0 | 0 | 6 | 0 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Redness, iNTS-GMMA full dose | 0 | 0 | 0 | 3 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Redness, TCV full dose | 0 | 0 | 0 | 0 | 0
  Redness, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Redness, Placebo | 0 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose | 4 | 0 | 0 | 0 | 0
  Pain, saline: number analyzed (Participants) | 4 | 0 | 15 | 0 | 10
  Pain, saline | 2 | 0 | 0 | 0 | 2
  Pain, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Pain, iNTS-GMMA low dose | 0 | 4 | 0 | 0 | 0
  Pain, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Pain, TCV low dose | 0 | 1 | 0 | 0 | 0
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 15 | 0 | 0
  Pain, iNTS-TCV full dose | 0 | 0 | 15 | 0 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Pain, iNTS-GMMA full dose | 0 | 0 | 0 | 14 | 0
  Pain, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Pain, TCV full dose | 0 | 0 | 0 | 7 | 0
  Pain, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Pain, Placebo | 0 | 0 | 0 | 0 | 5
  Swelling, iNTS-TCV Low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 07
  Swelling, iNTS-TCV Low dose | 0 | 0 | 0 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 4 | 0 | 15 | 0 | 10
  Swelling, saline | 0 | 0 | 0 | 0 | 0
  Swelling, TCV low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Swelling, TCV low dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 4 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 15 | 0 | 0
  Swelling, iNTS-TCV full dose | 0 | 0 | 2 | 0 | 0
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Swelling, TCV full dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 15 | 0
  Swelling, iNTS-GMMA full dose | 0 | 0 | 0 | 1 | 0
  Swelling, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Swelling, Placebo | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Stage 1: Number of Participants With Any Solicited Administration Site Events After the Third Study Intervention Administration
Description: as for outcome 14
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-third vaccination on Day 169)
Population: The analysis was performed on the Solicited safety set, which included all participants who received third dose of the study intervention and who had solicited safety data in the 7 days following third intervention. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 13 | 14 | 10
Participants
  Redness, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV low dose | 0 | 0 | 0 | 0 | 0
  Redness, Saline: number analyzed (Participants) | 4 | 0 | 13 | 0 | 10
  Redness, Saline | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Redness, iNTS-GMMA low dose | 0 | 0 | 0 | 0 | 0
  Redness, TCV low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Redness, TCV low dose | 0 | 0 | 0 | 0 | 0
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 13 | 0 | 0
  Redness, iNTS-TCV full dose | 0 | 0 | 3 | 0 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Redness, iNTS-GMMA full dose | 0 | 0 | 0 | 4 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Redness, TCV full dose | 0 | 0 | 0 | 4 | 0
  Redness, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Redness, Placebo | 0 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV low dose | 4 | 0 | 0 | 0 | 0
  Pain, saline: number analyzed (Participants) | 4 | 0 | 13 | 0 | 10
  Pain, saline | 1 | 0 | 1 | 0 | 1
  Pain, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Pain, iNTS-GMMA low dose | 0 | 3 | 0 | 0 | 0
  Pain, TCV low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Pain, TCV low dose | 0 | 0 | 0 | 0 | 0
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 13 | 0 | 0
  Pain, iNTS-TCV full dose | 0 | 0 | 11 | 0 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Pain, iNTS-GMMA full dose | 0 | 0 | 0 | 14 | 0
  Pain, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Pain, TCV full dose | 0 | 0 | 0 | 2 | 0
  Pain, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Pain, Placebo | 0 | 0 | 0 | 0 | 5
  Swelling, iNTS-TCV Low: number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
  Swelling, iNTS-TCV Low | 0 | 0 | 0 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 4 | 0 | 13 | 0 | 10
  Swelling, saline | 0 | 0 | 0 | 0 | 0
  Swelling, TCV low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Swelling, TCV low dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose: number analyzed (Participants) | 0 | 3 | 0 | 0 | 0
  Swelling, iNTS-GMMA low dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 0 | 0 | 13 | 0 | 0
  Swelling, iNTS-TCV full dose | 0 | 0 | 2 | 0 | 0
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Swelling, TCV full dose | 0 | 0 | 0 | 0 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Swelling, iNTS-GMMA full dose | 0 | 0 | 0 | 1 | 0
  Swelling, Placebo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10
  Swelling, Placebo | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Stage 1: Number of Participants With Any Solicited Systemic Events After the First Study Intervention Administration
Description: The solicited systemic events included arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain) and fever (pyrexia). Fever is defined as body temperature equal to or above (>=) 38.0 degrees Celsius (°C). The preferred location for measuring temperature is the axilla. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-first vaccination on Day 1)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants
  Arthralgia | 0 | 1 | 3 | 3 | 0
  Fatigue | 2 | 3 | 7 | 11 | 2
  Headache | 3 | 2 | 6 | 5 | 1
  Myalgia | 4 | 2 | 6 | 6 | 0
  Fever | 0 | 0 | 1 | 0 | 0

17. Primary Outcome: Stage 1: Number of Participants With Any Solicited Systemic Events After the Second Study Intervention Administration
Description: The solicited systemic events included arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain) and fever (pyrexia). Fever is defined as body temperature equal to or above (≥) 38.0 degrees Celsius (°C). The preferred location for measuring temperature is the axilla. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-second vaccination on Day 57)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 15 | 15 | 10
Participants
  Arthralgia | 1 | 0 | 1 | 2 | 0
  Fatigue | 2 | 1 | 7 | 6 | 1
  Headache | 1 | 1 | 5 | 6 | 0
  Myalgia | 2 | 0 | 4 | 4 | 1
  Fever | 0 | 1 | 2 | 1 | 0

18. Primary Outcome: Stage 1: Number of Participants With Any Solicited Systemic Events After the Third Study Intervention Administration
Description: as for outcome 17
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-third vaccination on Day 169)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 13 | 14 | 10
Participants
  Arthralgia | 0 | 1 | 1 | 2 | 0
  Fatigue | 0 | 1 | 4 | 7 | 0
  Headache | 0 | 1 | 3 | 7 | 3
  Myalgia | 1 | 1 | 5 | 10 | 0
  Fever | 0 | 0 | 1 | 1 | 0

19. Primary Outcome: Stage 1: Number of Participants With Any Unsolicited Adverse Events (AE) After the First Study Intervention Administration
Description: An unsolicited AE is an AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited AE. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-first vaccination on Day 1)
Population: The analysis was performed on the unsolicited safety set, which included all participants who received the first dose of the study intervention and reported having/not having unsolicited AEs during the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants | 4 | 2 | 14 | 13 | 4

20. Primary Outcome: Stage 1: Number of Participants With Any Unsolicited AEs After the Second Study Intervention Administration
Description: as for outcome 19
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-second vaccination on Day 57)
Population: The analysis was performed on the unsolicited safety set, which included all participants who received the second dose of the study intervention and reported having/not having unsolicited AEs during the specified timepoints. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 15 | 15 | 10
Participants | 3 | 1 | 8 | 8 | 2

21. Primary Outcome: Stage 1: Number of Participants With Any Unsolicited AEs After the Third Study Intervention Administration
Description: as for outcome 19
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-third vaccination on Day 169)
Population: The analysis was performed on the unsolicited safety set, which included all participants who received the third dose of the study intervention and reported having/not having unsolicited AEs during the specified timepoints. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 13 | 14 | 10
Participants | 0 | 1 | 3 | 5 | 5

22. Primary Outcome: Stage 1: Number of Participants With Any Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From first study intervention administration (Day 1) up to 28 days after the third study intervention administration (Day 197)
Population: The analysis was performed on the exposed set, which included all participants who received at least 1 dose of the study intervention. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants | 0 | 0 | 0 | 1 | 0

23. Primary Outcome: Stage 1: Number of Participants With Any AEs/SAEs Leading to Withdrawal From the Study
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement. An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact. Any = occurrence of the event regardless of intensity grade.
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants | 0 | 0 | 0 | 0 | 0

24. Primary Outcome: Stage 1: Number of Participants With Any AEs/SAEs Leading to Withholding Further Study Intervention Administration
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
  An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention.
  AEs/SAEs that lead to withholding of the study intervention administration were considered under this outcome measure. Any = occurrence of the event regardless of intensity grade.
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants | 0 | 0 | 1 | 1 | 0

25. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 8
Description: Assessed hepatic laboratory parameters included alanine aminotransferase [ALT] and aspartate aminotransferase [AST], and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 1 (baseline) and Day 8 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 8)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 8 (7 days after the first study intervention administration) compared to Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants
  ALT: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 8) | 4 | 4 | 13 | 16 | 10
  ALT: Above (baseline) - within (Day 8) | 0 | 0 | 1 | 0 | 0
  ALT: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - above (Day 8) | 0 | 0 | 2 | 0 | 0
  AST: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 8) | 3 | 4 | 14 | 16 | 9
  AST: Above (baseline) - within (Day 8) | 1 | 0 | 0 | 0 | 1
  AST: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - above (Day 8) | 0 | 0 | 2 | 0 | 0
  Creatinine: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 8) | 2 | 3 | 14 | 13 | 8
  Creatinine: Above (baseline) - within (Day 8) | 1 | 0 | 0 | 1 | 0
  Creatinine: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 8) | 0 | 1 | 1 | 1 | 2
  Creatinine: Above (baseline) - above (Day 8) | 1 | 0 | 1 | 1 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 8) | 0 | 0 | 1 | 1 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 8) | 4 | 4 | 15 | 15 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 8) | 4 | 4 | 16 | 16 | 10
  Basophils: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 8) | 4 | 4 | 15 | 16 | 10
  Eosinophils: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 8) | 0 | 0 | 1 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 8) | 4 | 4 | 16 | 16 | 9
  Hemoglobin: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 8) | 4 | 4 | 15 | 15 | 10
  Lymphocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 8) | 0 | 0 | 1 | 0 | 0
  Monocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 8) | 4 | 4 | 15 | 16 | 10
  Monocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 8) | 0 | 0 | 1 | 0 | 0
  Monocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 8) | 3 | 4 | 12 | 15 | 9
  Neutrophils: Above (baseline) - within (Day 8) | 1 | 0 | 3 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 8) | 0 | 0 | 1 | 0 | 1
  Neutrophils: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 8) | 0 | 1 | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 8) | 3 | 3 | 11 | 15 | 10
  Platelets: Above (baseline) - within (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 8) | 0 | 0 | 5 | 1 | 0
  Platelets: Above (baseline) - above (Day 8) | 1 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - below (Day 8) | 0 | 2 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 1
  White Blood Cells [WBC]: Above (baseline) - below (Day 8) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 8) | 1 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 8) | 3 | 2 | 15 | 16 | 9
  White Blood Cells [WBC]: Above (baseline) - within (Day 8) | 0 | 0 | 1 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 8) | 0 | 0 | 0 | 0 | 0

26. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 64
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 57 (baseline) and Day 64 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 64)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 64 (7 days after the second study intervention administration) compared to Baseline (Day 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 15 | 15 | 10
Participants
  ALT: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 64) | 4 | 4 | 12 | 14 | 10
  ALT: Above (baseline) - within (Day 64) | 0 | 0 | 2 | 0 | 0
  ALT: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 1 | 0
  ALT: Above (baseline) - above (Day 64) | 0 | 0 | 1 | 0 | 0
  AST: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 64) | 2 | 4 | 13 | 14 | 10
  AST: Above (baseline) - within (Day 64) | 1 | 0 | 1 | 1 | 0
  AST: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 64) | 1 | 0 | 0 | 0 | 0
  AST: Above (baseline) - above (Day 64) | 0 | 0 | 1 | 0 | 0
  Creatinine: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 64) | 3 | 4 | 14 | 13 | 7
  Creatinine: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 1 | 2
  Creatinine: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 1
  Creatinine: Above (baseline) - above (Day 64) | 1 | 0 | 1 | 1 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 64) | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 64) | 3 | 4 | 15 | 14 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 1 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 64) | 4 | 4 | 15 | 15 | 10
  Basophils: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 64) | 4 | 4 | 15 | 15 | 10
  Eosinophils: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 1
  Hemoglobin: Within (baseline) - within (Day 64) | 4 | 4 | 15 | 15 | 9
  Hemoglobin: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 64) | 4 | 4 | 15 | 15 | 9
  Lymphocytes: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 64) | 4 | 4 | 15 | 15 | 10
  Monocytes: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 64) | 3 | 4 | 11 | 14 | 6
  Neutrophils: Above (baseline) - within (Day 64) | 0 | 0 | 1 | 1 | 2
  Neutrophils: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 64) | 1 | 0 | 2 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 64) | 0 | 0 | 1 | 0 | 2
  Platelets: Below (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 64) | 0 | 1 | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 64) | 3 | 3 | 13 | 13 | 10
  Platelets: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 64) | 0 | 0 | 1 | 2 | 0
  Platelets: Above (baseline) - above (Day 64) | 1 | 0 | 1 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - below (Day 64) | 0 | 1 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 64) | 1 | 0 | 1 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 64) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 64) | 3 | 3 | 14 | 15 | 7
  White Blood Cells [WBC]: Above (baseline) - within (Day 64) | 0 | 0 | 0 | 0 | 2
  White Blood Cells [WBC]: Below (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 64) | 0 | 0 | 0 | 0 | 1

27. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 176
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 169 (baseline) and Day 176 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 176)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 176 (7 days after the third study intervention administration) compared to Baseline (Day 169)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 13 | 14 | 10
Participants
  ALT: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 176) | 4 | 3 | 11 | 13 | 10
  ALT: Above (baseline) - within (Day 176) | 0 | 0 | 1 | 0 | 0
  ALT: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 176) | 0 | 0 | 1 | 1 | 0
  ALT: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 176) | 4 | 3 | 12 | 14 | 10
  AST: Above (baseline) - within (Day 176) | 0 | 0 | 1 | 0 | 0
  AST: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 176) | 3 | 3 | 10 | 10 | 6
  Creatinine: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 1
  Creatinine: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 176) | 0 | 0 | 2 | 3 | 2
  Creatinine: Above (baseline) - above (Day 176) | 1 | 0 | 1 | 1 | 1
  Blood Urea Nitrogen: Below (baseline) - below (Day 176) | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 176) | 3 | 3 | 13 | 13 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 1 | 0
  Basophils: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 176) | 4 | 3 | 13 | 14 | 10
  Basophils: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 176) | 4 | 3 | 12 | 14 | 10
  Eosinophils: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 176) | 0 | 0 | 1 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 1 | 0
  Hemoglobin: Within (baseline) - within (Day 176) | 4 | 3 | 13 | 13 | 9
  Hemoglobin: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 176) | 4 | 3 | 13 | 14 | 10
  Lymphocytes: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 176) | 4 | 3 | 13 | 14 | 10
  Monocytes: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 176) | 1 | 3 | 8 | 11 | 8
  Neutrophils: Above (baseline) - within (Day 176) | 1 | 0 | 2 | 1 | 1
  Neutrophils: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 176) | 2 | 0 | 2 | 1 | 1
  Neutrophils: Above (baseline) - above (Day 176) | 0 | 0 | 1 | 1 | 0
  Platelets: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 176) | 2 | 3 | 9 | 12 | 10
  Platelets: Above (baseline) - within (Day 176) | 0 | 0 | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 176) | 2 | 0 | 2 | 1 | 0
  Platelets: Above (baseline) - above (Day 176) | 0 | 0 | 1 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 176) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 176) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 176) | 4 | 3 | 13 | 12 | 9
  White Blood Cells [WBC]: Above (baseline) - within (Day 176) | 0 | 0 | 0 | 1 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 176) | 0 | 0 | 0 | 1 | 1
  White Blood Cells [WBC]: Above (baseline) - above (Day 176) | 0 | 0 | 0 | 0 | 0

28. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 29
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 1 (baseline) and Day 29 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 29)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 29 (28 days after the first study intervention administration) compared to Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 10
Participants
  ALT: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 29) | 4 | 4 | 13 | 16 | 10
  ALT: Above (baseline) - within (Day 29) | 0 | 0 | 1 | 0 | 0
  ALT: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - above (Day 29) | 0 | 0 | 2 | 0 | 0
  AST: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 29) | 3 | 4 | 14 | 16 | 9
  AST: Above (baseline) - within (Day 29) | 1 | 0 | 2 | 0 | 1
  AST: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 29) | 2 | 4 | 15 | 14 | 8
  Creatinine: Above (baseline) - within (Day 29) | 1 | 0 | 0 | 2 | 0
  Creatinine: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 2
  Creatinine: Above (baseline) - above (Day 29) | 1 | 0 | 1 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 29) | 0 | 0 | 1 | 1 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 29) | 4 | 4 | 15 | 15 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 29) | 4 | 4 | 16 | 16 | 10
  Basophils: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 29) | 4 | 4 | 15 | 16 | 10
  Eosinophils: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 29) | 0 | 0 | 1 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 29) | 4 | 4 | 16 | 15 | 9
  Hemoglobin: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 1 | 0
  Hemoglobin: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 29) | 4 | 4 | 15 | 16 | 10
  Lymphocytes: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 29) | 0 | 0 | 1 | 0 | 0
  Monocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 29) | 4 | 4 | 16 | 15 | 10
  Monocytes: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 29) | 0 | 0 | 0 | 1 | 0
  Monocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 29) | 3 | 4 | 12 | 14 | 9
  Neutrophils: Above (baseline) - within (Day 29) | 0 | 0 | 1 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 29) | 0 | 0 | 1 | 1 | 1
  Neutrophils: Above (baseline) - above (Day 29) | 1 | 0 | 2 | 0 | 0
  Platelets: Below (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 29) | 0 | 1 | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 29) | 2 | 3 | 14 | 16 | 10
  Platelets: Above (baseline) - within (Day 29) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 29) | 1 | 0 | 2 | 0 | 0
  Platelets: Above (baseline) - above (Day 29) | 1 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - below (Day 29) | 0 | 1 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 29) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 29) | 1 | 1 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 29) | 3 | 2 | 14 | 15 | 10
  White Blood Cells [WBC]: Above (baseline) - within (Day 29) | 0 | 0 | 1 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 29) | 0 | 0 | 1 | 1 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 29) | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 85
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 57 (baseline) and Day 85 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 85)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 85 (28 days after the second study intervention administration) compared to Baseline (Day 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 4 | 15 | 15 | 10
Participants
  ALT: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 85) | 4 | 4 | 11 | 15 | 10
  ALT: Above (baseline) - within (Day 85) | 0 | 0 | 2 | 0 | 0
  ALT: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 85) | 0 | 0 | 1 | 0 | 0
  ALT: Above (baseline) - above (Day 85) | 0 | 0 | 1 | 0 | 0
  AST: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 85) | 3 | 4 | 13 | 13 | 10
  AST: Above (baseline) - within (Day 85) | 1 | 0 | 2 | 1 | 0
  AST: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 1 | 0
  AST: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 85) | 3 | 4 | 12 | 11 | 7
  Creatinine: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 1
  Creatinine: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 85) | 0 | 0 | 2 | 2 | 1
  Creatinine: Above (baseline) - above (Day 85) | 1 | 0 | 1 | 2 | 1
  Blood Urea Nitrogen: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 85) | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 85) | 3 | 4 | 15 | 15 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 85) | 4 | 4 | 15 | 15 | 10
  Basophils: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 85) | 4 | 4 | 15 | 15 | 10
  Eosinophils: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 1
  Hemoglobin: Within (baseline) - within (Day 85) | 4 | 4 | 15 | 14 | 9
  Hemoglobin: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 85) | 4 | 4 | 15 | 14 | 10
  Lymphocytes: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 85) | 4 | 4 | 15 | 15 | 10
  Monocytes: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 85) | 4 | 4 | 13 | 14 | 6
  Neutrophils: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 4
  Neutrophils: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 85) | 0 | 0 | 2 | 1 | 0
  Platelets: Below (baseline) - below (Day 85) | 0 | 1 | 0 | 0 | 0
  Platelets: Within (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 85) | 3 | 3 | 13 | 15 | 10
  Platelets: Above (baseline) - within (Day 85) | 0 | 0 | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 85) | 0 | 0 | 1 | 0 | 0
  Platelets: Above (baseline) - above (Day 85) | 1 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - below (Day 85) | 0 | 1 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 85) | 0 | 1 | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 85) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 85) | 4 | 2 | 15 | 14 | 7
  White Blood Cells [WBC]: Above (baseline) - within (Day 85) | 0 | 0 | 0 | 0 | 3
  White Blood Cells [WBC]: Below (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 85) | 0 | 0 | 0 | 1 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 85) | 0 | 0 | 0 | 0 | 0

30. Primary Outcome: Stage 1: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 197
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 169 (baseline) and Day 197 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 197)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 197 (28 days after the third study intervention administration) compared to Baseline (Day 169)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group
Number analyzed (Participants) | 4 | 3 | 13 | 14 | 10
Participants
  ALT: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 197) | 4 | 3 | 10 | 14 | 10
  ALT: Above (baseline) - within (Day 197) | 0 | 0 | 1 | 0 | 0
  ALT: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 197) | 0 | 0 | 2 | 0 | 0
  ALT: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - within (Day 197) | 4 | 3 | 12 | 13 | 10
  AST: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  AST: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 1 | 0
  AST: Above (baseline) - above (Day 197) | 0 | 0 | 1 | 0 | 0
  Creatinine: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 197) | 2 | 3 | 11 | 13 | 7
  Creatinine: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 197) | 1 | 0 | 1 | 0 | 1
  Creatinine: Above (baseline) - above (Day 197) | 1 | 0 | 1 | 1 | 2
  Blood Urea Nitrogen: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 197) | 1 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - within (Day 197) | 3 | 3 | 13 | 13 | 10
  Blood Urea Nitrogen: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 1 | 0
  Basophils: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 197) | 4 | 3 | 13 | 14 | 10
  Basophils: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 197) | 4 | 3 | 13 | 14 | 10
  Eosinophils: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 197) | 0 | 0 | 1 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 197) | 4 | 3 | 11 | 12 | 9
  Hemoglobin: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 197) | 0 | 0 | 1 | 1 | 0
  Hemoglobin: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 197) | 4 | 3 | 13 | 13 | 10
  Lymphocytes: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 1 | 0
  Lymphocytes: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 197) | 4 | 3 | 13 | 14 | 10
  Monocytes: Above (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 197) | 0 | 0 | 1 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 197) | 3 | 3 | 9 | 11 | 9
  Neutrophils: Above (baseline) - within (Day 197) | 1 | 0 | 2 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 197) | 0 | 0 | 0 | 1 | 0
  Neutrophils: Above (baseline) - above (Day 197) | 0 | 0 | 1 | 1 | 1
  Platelets: Below (baseline) - below (Day 197) | 0 | 0 | 0 | 1 | 0
  Platelets: Within (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 197) | 3 | 2 | 11 | 13 | 10
  Platelets: Above (baseline) - within (Day 197) | 0 | 0 | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 197) | 1 | 1 | 0 | 0 | 0
  Platelets: Above (baseline) - above (Day 197) | 0 | 0 | 1 | 0 | 0
  White Blood Cells (WBC): Below (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  White Blood Cells (WBC): Within (baseline) - below (Day 197) | 0 | 1 | 1 | 0 | 0
  White Blood Cells (WBC): Above (baseline) - below (Day 197) | 0 | 0 | 0 | 0 | 0
  White Blood Cells (WBC): Below (baseline) - within (Day 197) | 0 | 0 | 0 | 0 | 0
  White Blood Cells (WBC): Within (baseline) - within (Day 197) | 4 | 2 | 12 | 12 | 10
  White Blood Cells (WBC): Above (baseline) - within (Day 197) | 0 | 0 | 0 | 1 | 0
  White Blood Cells (WBC): Below (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0
  White Blood Cells (WBC): Within (baseline) - above (Day 197) | 0 | 0 | 0 | 1 | 0
  White Blood Cells (WBC): Above (baseline) - above (Day 197) | 0 | 0 | 0 | 0 | 0

31. Primary Outcome: Stage 2: Number of Participants With Any Solicited Administration Site Events After the First Study Intervention Administration
Description: as for outcome 14
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-first vaccination on Day 1)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Redness, iNTS-TCV full dose | 2 | 0 | 0
  Redness, saline: number analyzed (Participants) | 45 | 0 | 15
  Redness, saline | 0 | 0 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 45 | 0
  Redness, TCV full dose | 0 | 3 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 45 | 0
  Redness, iNTS-GMMA full dose | 0 | 7 | 0
  Redness, control: number analyzed (Participants) | 0 | 0 | 15
  Redness, control | 0 | 0 | 0
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Pain, iNTS-TCV full dose | 38 | 0 | 0
  Pain, saline: number analyzed (Participants) | 45 | 0 | 15
  Pain, saline | 16 | 0 | 5
  Pain, TCV full dose: number analyzed (Participants) | 0 | 45 | 0
  Pain, TCV full dose | 0 | 20 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 45 | 0
  Pain, iNTS-GMMA full dose | 0 | 41 | 0
  Pain, control: number analyzed (Participants) | 0 | 0 | 15
  Pain, control | 0 | 0 | 6
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Swelling, iNTS-TCV full dose | 7 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 45 | 0 | 15
  Swelling, saline | 1 | 0 | 0
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 45 | 0
  Swelling, TCV full dose | 0 | 2 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 45 | 0
  Swelling, iNTS-GMMA full dose | 0 | 10 | 0
  Swelling, control: number analyzed (Participants) | 0 | 0 | 15
  Swelling, control | 0 | 0 | 0

32. Primary Outcome: Stage 2: Number of Participants With Any Solicited Administration Site Events After the Second Study Intervention Administration
Description: as for outcome 14
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-second vaccination on Day 57)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 43 | 15
Participants
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Redness, iNTS-TCV full dose | 1 | 0 | 0
  Redness, saline: number analyzed (Participants) | 45 | 0 | 15
  Redness, saline | 1 | 0 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 43 | 0
  Redness, TCV full dose | 0 | 2 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 43 | 0
  Redness, iNTS-GMMA full dose | 0 | 3 | 0
  Redness, control: number analyzed (Participants) | 0 | 0 | 15
  Redness, control | 0 | 0 | 1
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Pain, iNTS-TCV full dose | 35 | 0 | 0
  Pain, saline: number analyzed (Participants) | 45 | 0 | 15
  Pain, saline | 14 | 0 | 5
  Pain, TCV full dose: number analyzed (Participants) | 0 | 43 | 0
  Pain, TCV full dose | 0 | 24 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 43 | 0
  Pain, iNTS-GMMA full dose | 0 | 41 | 0
  Pain, control: number analyzed (Participants) | 0 | 0 | 15
  Pain, control | 0 | 0 | 9
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 45 | 0 | 0
  Swelling, iNTS-TCV full dose | 6 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 45 | 0 | 15
  Swelling, saline | 2 | 0 | 0
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 43 | 0
  Swelling, TCV full dose | 0 | 6 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 43 | 0
  Swelling, iNTS-GMMA full dose | 0 | 11 | 0
  Swelling, control: number analyzed (Participants) | 0 | 0 | 15
  Swelling, control | 0 | 0 | 2

33. Primary Outcome: Stage 2: Number of Participants With Any Solicited Administration Site Events After the Third Study Intervention Administration
Description: as for outcome 14
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-third vaccination on Day 169)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 42 | 38 | 14
Participants
  Redness, iNTS-TCV full dose: number analyzed (Participants) | 42 | 0 | 0
  Redness, iNTS-TCV full dose | 4 | 0 | 0
  Redness, saline: number analyzed (Participants) | 42 | 0 | 14
  Redness, saline | 0 | 0 | 0
  Redness, TCV full dose: number analyzed (Participants) | 0 | 38 | 0
  Redness, TCV full dose | 0 | 1 | 0
  Redness, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 38 | 0
  Redness, iNTS-GMMA full dose | 0 | 3 | 0
  Redness, control: number analyzed (Participants) | 0 | 0 | 14
  Redness, control | 0 | 0 | 0
  Pain, iNTS-TCV full dose: number analyzed (Participants) | 42 | 0 | 0
  Pain, iNTS-TCV full dose | 32 | 0 | 0
  Pain, saline: number analyzed (Participants) | 42 | 0 | 14
  Pain, saline | 10 | 0 | 6
  Pain, TCV full dose: number analyzed (Participants) | 0 | 38 | 0
  Pain, TCV full dose | 0 | 19 | 0
  Pain, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 38 | 0
  Pain, iNTS-GMMA full dose | 0 | 35 | 0
  Pain, control: number analyzed (Participants) | 0 | 0 | 14
  Pain, control | 0 | 0 | 8
  Swelling, iNTS-TCV full dose: number analyzed (Participants) | 42 | 0 | 0
  Swelling, iNTS-TCV full dose | 5 | 0 | 0
  Swelling, saline: number analyzed (Participants) | 42 | 0 | 14
  Swelling, saline | 2 | 0 | 1
  Swelling, TCV full dose: number analyzed (Participants) | 0 | 38 | 0
  Swelling, TCV full dose | 0 | 2 | 0
  Swelling, iNTS-GMMA full dose: number analyzed (Participants) | 0 | 38 | 0
  Swelling, iNTS-GMMA full dose | 0 | 9 | 0
  Swelling, control: number analyzed (Participants) | 0 | 0 | 14
  Swelling, control | 0 | 0 | 1

34. Primary Outcome: Stage 2: Number of Participants With Any Solicited Systemic Events After the First Study Intervention Administration
Description: The solicited systemic events included arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain) and fever (pyrexia). Fever is defined as body temperature >=38.0 degrees Celsius (°C). The preferred location for measuring temperature is the axilla. Any = occurrence of the event regardless of intensity grade.
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-first vaccination on Day 1)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants
  Arthralgia | 12 | 10 | 3
  Fatigue | 23 | 20 | 4
  Headache | 26 | 24 | 5
  Myalgia | 23 | 21 | 3
  Fever | 8 | 6 | 0

35. Primary Outcome: Stage 2: Number of Participants With Solicited Systemic Events After the Second Study Intervention Administration
Description: as for outcome 34
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-second vaccination on Day 57)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 43 | 15
Participants
  Arthralgia | 11 | 11 | 5
  Fatigue | 18 | 24 | 4
  Headache | 22 | 26 | 5
  Myalgia | 18 | 20 | 5
  Fever | 5 | 5 | 0

36. Primary Outcome: Stage 2: Number of Participants With Any Solicited Systemic Events After the Third Study Intervention Administration
Description: as for outcome 34
Time Frame: Within 7 days post vaccination (day of administration and 6 subsequent days post-third vaccination on Day 169)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 42 | 38 | 14
Participants
  Arthralgia | 13 | 15 | 3
  Fatigue | 18 | 18 | 2
  Headache | 21 | 23 | 2
  Myalgia | 17 | 18 | 4
  Fever | 4 | 9 | 0

37. Primary Outcome: Stage 2: Number of Participants With Any Unsolicited AE After the First Study Intervention Administration
Description: as for outcome 19
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-first vaccination on Day 1)
Population: The analysis was performed on the unsolicited safety set, which included all participants who received the first dose of the study intervention and reported having/not having unsolicited AEs during the specified timepoints. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants | 21 | 24 | 8

38. Primary Outcome: Stage 2: Number of Participants With Any Unsolicited AE After the Second Study Intervention Administration
Description: as for outcome 19
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-second vaccination on Day 57)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 43 | 15
Participants | 13 | 17 | 3

39. Primary Outcome: Stage 2: Number of Participants With Any Unsolicited AE After the Third Study Intervention Administration
Description: as for outcome 19
Time Frame: Within 28 days post vaccination (day of administration and 27 subsequent days post-third vaccination on Day 169)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 42 | 38 | 14
Participants | 13 | 12 | 1

40. Primary Outcome: Stage 2: Number of Participants With Any SAEs
Description: as for outcome 1
Time Frame: as for outcome 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants | 0 | 1 | 0

41. Primary Outcome: Stage 2: Number of Participants With Any AEs/SAEs Leading to Withdrawal From the Study
Description: as for outcome 2
Time Frame: From first study intervention administration (Day 1) up to 28 days after the third study intervention (Day 197)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants | 0 | 0 | 0

42. Primary Outcome: Stage 2: Number of Participants With Any AEs/SAEs Leading to Withholding Further Study Intervention Administration
Description: AEs/SAEs that lead to withholding of the study intervention administration were considered under this outcome measure. Any = occurrence of the event regardless of intensity grade.
Time Frame: From first study intervention administration (Day 1) up to 28 days after the third study intervention (Day 197)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants | 0 | 0 | 0

43. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 8
Description: Assessed hepatic laboratory parameters included ALT and AST, and renal laboratory parameters included creatinine and urea/blood urea nitrogen. Hematological laboratory parameters included basophils, eosinophils, hemoglobin, lymphocytes, monocytes, neutrophils, platelets and white blood cells (WBCs). Categories reported when comparing Day 1 (baseline) and Day 8 hematological, renal and hepatic laboratory results are defined as follows: <range> (at baseline) - <range> (at timing) (e.g. Within (Baseline) - Within (Day 8)) where range is being classified as below, within or above the normal range. Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: At Day 8 (7 days after the first study intervention administration) compared to Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants
  ALT: Below (baseline) - below (Day 8) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 8) | 2 | 1 | 0
  ALT: Above (baseline) - below (Day 8) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 8) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 8) | 36 | 35 | 13
  ALT: Above (baseline) - within (Day 8) | 3 | 5 | 2
  ALT: Below (baseline) - above (Day 8) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 8) | 2 | 2 | 0
  ALT: Above (baseline) - above (Day 8) | 2 | 2 | 0
  AST: Below (baseline) - below (Day 8) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 8) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 8) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 8) | 1 | 0 | 0
  AST: Within (baseline) - within (Day 8) | 37 | 43 | 12
  AST: Above (baseline) - within (Day 8) | 2 | 2 | 3
  AST: Below (baseline) - above (Day 8) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 8) | 3 | 0 | 0
  AST: Above (baseline) - above (Day 8) | 2 | 0 | 0
  Creatinine: Below (baseline) - below (Day 8) | 2 | 3 | 0
  Creatinine: Within (baseline) - below (Day 8) | 1 | 1 | 1
  Creatinine: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 8) | 1 | 0 | 1
  Creatinine: Within (baseline) - within (Day 8) | 41 | 41 | 13
  Creatinine: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 8) | 6 | 5 | 1
  Blood Urea Nitrogen: Within (baseline) - below (Day 8) | 11 | 4 | 0
  Blood Urea Nitrogen: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 8) | 6 | 7 | 3
  Blood Urea Nitrogen: Within (baseline) - within (Day 8) | 22 | 29 | 11
  Blood Urea Nitrogen: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 8) | 45 | 44 | 15
  Basophils: Above (baseline) - within (Day 8) | 0 | 1 | 0
  Basophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 8) | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 8) | 44 | 45 | 15
  Eosinophils: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 8) | 1 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 8) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 8) | 1 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 8) | 38 | 39 | 11
  Hemoglobin: Above (baseline) - within (Day 8) | 1 | 2 | 0
  Hemoglobin: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 8) | 1 | 1 | 2
  Hemoglobin: Above (baseline) - above (Day 8) | 3 | 2 | 2
  Lymphocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 8) | 43 | 43 | 13
  Lymphocytes: Above (baseline) - within (Day 8) | 0 | 0 | 2
  Lymphocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 8) | 1 | 2 | 0
  Lymphocytes: Above (baseline) - above (Day 8) | 1 | 0 | 0
  Monocytes: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 8) | 39 | 44 | 15
  Monocytes: Above (baseline) - within (Day 8) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 8) | 6 | 1 | 0
  Monocytes: Above (baseline) - above (Day 8) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 8) | 41 | 42 | 15
  Neutrophils: Above (baseline) - within (Day 8) | 1 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 8) | 3 | 1 | 0
  Neutrophils: Above (baseline) - above (Day 8) | 0 | 1 | 0
  Platelets: Below (baseline) - below (Day 8) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 8) | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 8) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 8) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 8) | 35 | 32 | 11
  Platelets: Above (baseline) - within (Day 8) | 0 | 1 | 1
  Platelets: Below (baseline) - above (Day 8) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 8) | 5 | 5 | 1
  Platelets: Above (baseline) - above (Day 8) | 4 | 6 | 2
  White Blood Cells [WBC]: Below (baseline) - below (Day 8) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 8) | 0 | 1 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 8) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 8) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 8) | 41 | 41 | 14
  White Blood Cells [WBC]: Above (baseline) - within (Day 8) | 0 | 2 | 1
  White Blood Cells [WBC]: Below (baseline) - above (Day 8) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 8) | 3 | 1 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 8) | 1 | 0 | 0

44. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 64
Description: as for outcome 26
Time Frame: At Day 64 (7 days after the second study intervention administration) compared to Baseline (Day 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 43 | 15
Participants
  ALT: Below (baseline) - below (Day 64) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 64) | 1 | 1 | 0
  ALT: Above (baseline) - below (Day 64) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 64) | 1 | 0 | 0
  ALT: Within (baseline) - within (Day 64) | 38 | 35 | 12
  ALT: Above (baseline) - within (Day 64) | 2 | 4 | 0
  ALT: Below (baseline) - above (Day 64) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 64) | 2 | 1 | 1
  ALT: Above (baseline) - above (Day 64) | 1 | 2 | 2
  AST: Below (baseline) - below (Day 64) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 64) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 64) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 64) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 64) | 40 | 39 | 11
  AST: Above (baseline) - within (Day 64) | 1 | 4 | 0
  AST: Below (baseline) - above (Day 64) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 64) | 1 | 0 | 1
  AST: Above (baseline) - above (Day 64) | 3 | 0 | 3
  Creatinine: Below (baseline) - below (Day 64) | 3 | 3 | 0
  Creatinine: Within (baseline) - below (Day 64) | 1 | 2 | 0
  Creatinine: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 64) | 0 | 4 | 1
  Creatinine: Within (baseline) - within (Day 64) | 41 | 34 | 14
  Creatinine: Above (baseline) - within (Day 64) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 64) | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 64) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 64) | 6 | 5 | 4
  Blood Urea Nitrogen: Within (baseline) - below (Day 64) | 4 | 8 | 1
  Blood Urea Nitrogen: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 64) | 9 | 2 | 2
  Blood Urea Nitrogen: Within (baseline) - within (Day 64) | 26 | 28 | 8
  Blood Urea Nitrogen: Above (baseline) - within (Day 64) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 64) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 64) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 64) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 64) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 64) | 44 | 43 | 15
  Basophils: Above (baseline) - within (Day 64) | 1 | 0 | 0
  Basophils: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 64) | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 64) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 64) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 64) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 64) | 40 | 43 | 15
  Eosinophils: Above (baseline) - within (Day 64) | 1 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 64) | 1 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 64) | 3 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 64) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 64) | 0 | 1 | 0
  Hemoglobin: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 64) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 64) | 37 | 37 | 13
  Hemoglobin: Above (baseline) - within (Day 64) | 1 | 2 | 0
  Hemoglobin: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 64) | 1 | 0 | 0
  Hemoglobin: Above (baseline) - above (Day 64) | 4 | 3 | 2
  Lymphocytes: Below (baseline) - below (Day 64) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 64) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 64) | 43 | 42 | 15
  Lymphocytes: Above (baseline) - within (Day 64) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 64) | 2 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 64) | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 64) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 64) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 64) | 44 | 41 | 15
  Monocytes: Above (baseline) - within (Day 64) | 1 | 1 | 0
  Monocytes: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 64) | 0 | 1 | 0
  Monocytes: Above (baseline) - above (Day 64) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 64) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 64) | 0 | 1 | 0
  Neutrophils: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 64) | 41 | 39 | 15
  Neutrophils: Above (baseline) - within (Day 64) | 2 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 64) | 1 | 1 | 0
  Neutrophils: Above (baseline) - above (Day 64) | 1 | 1 | 0
  Platelets: Below (baseline) - below (Day 64) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 64) | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 64) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 64) | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 64) | 34 | 35 | 12
  Platelets: Above (baseline) - within (Day 64) | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 64) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 64) | 3 | 3 | 0
  Platelets: Above (baseline) - above (Day 64) | 6 | 5 | 3
  White Blood Cells [WBC]: Below (baseline) - below (Day 64) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 64) | 1 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 64) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 64) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 64) | 40 | 41 | 15
  White Blood Cells [WBC]: Above (baseline) - within (Day 64) | 2 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 64) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 64) | 1 | 2 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 64) | 1 | 0 | 0

45. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 176
Description: as for outcome 27
Time Frame: At Day 176 (7 days after the third study intervention administration) compared to Baseline (Day 169)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 42 | 38 | 14
Participants
  ALT: Below (baseline) - below (Day 176) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 176) | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 176) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 176) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 176) | 37 | 34 | 14
  ALT: Above (baseline) - within (Day 176) | 3 | 2 | 0
  ALT: Below (baseline) - above (Day 176) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 176) | 1 | 2 | 0
  ALT: Above (baseline) - above (Day 176) | 1 | 0 | 0
  AST: Below (baseline) - below (Day 176) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 176) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 176) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 176) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 176) | 34 | 33 | 13
  AST: Above (baseline) - within (Day 176) | 3 | 3 | 0
  AST: Below (baseline) - above (Day 176) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 176) | 3 | 1 | 0
  AST: Above (baseline) - above (Day 176) | 2 | 1 | 1
  Creatinine: Below (baseline) - below (Day 176) | 4 | 3 | 1
  Creatinine: Within (baseline) - below (Day 176) | 3 | 1 | 0
  Creatinine: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 176) | 0 | 1 | 0
  Creatinine: Within (baseline) - within (Day 176) | 35 | 33 | 13
  Creatinine: Above (baseline) - within (Day 176) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 176) | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 176) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 176) | 5 | 5 | 2
  Blood Urea Nitrogen: Within (baseline) - below (Day 176) | 7 | 5 | 5
  Blood Urea Nitrogen: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 176) | 7 | 0 | 2
  Blood Urea Nitrogen: Within (baseline) - within (Day 176) | 23 | 28 | 5
  Blood Urea Nitrogen: Above (baseline) - within (Day 176) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 176) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 176) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 176) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 176) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 176) | 42 | 38 | 14
  Basophils: Above (baseline) - within (Day 176) | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 176) | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 176) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 176) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 176) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 176) | 42 | 38 | 14
  Eosinophils: Above (baseline) - within (Day 176) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 176) | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 176) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 176) | 2 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 176) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 176) | 25 | 28 | 7
  Hemoglobin: Above (baseline) - within (Day 176) | 5 | 4 | 3
  Hemoglobin: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 176) | 4 | 2 | 0
  Hemoglobin: Above (baseline) - above (Day 176) | 6 | 4 | 4
  Lymphocytes: Below (baseline) - below (Day 176) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 176) | 0 | 0 | 14
  Lymphocytes: Within (baseline) - within (Day 176) | 40 | 36 | 0
  Lymphocytes: Above (baseline) - within (Day 176) | 1 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 176) | 0 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 176) | 1 | 1 | 0
  Monocytes: Below (baseline) - below (Day 176) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 176) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 176) | 39 | 37 | 14
  Monocytes: Above (baseline) - within (Day 176) | 1 | 1 | 0
  Monocytes: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 176) | 1 | 0 | 0
  Monocytes: Above (baseline) - above (Day 176) | 1 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 176) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 176) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 176) | 40 | 35 | 14
  Neutrophils: Above (baseline) - within (Day 176) | 0 | 0 | 0
  Neutrophils: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 176) | 2 | 1 | 0
  Neutrophils: Above (baseline) - above (Day 176) | 0 | 2 | 0
  Platelets: Below (baseline) - below (Day 176) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 176) | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 176) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 176) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 176) | 29 | 24 | 11
  Platelets: Above (baseline) - within (Day 176) | 1 | 0 | 0
  Platelets: Below (baseline) - above (Day 176) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 176) | 6 | 4 | 1
  Platelets: Above (baseline) - above (Day 176) | 5 | 9 | 2
  White Blood Cells [WBC]: Below (baseline) - below (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 176) | 41 | 36 | 14
  White Blood Cells [WBC]: Above (baseline) - within (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 176) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 176) | 1 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 176) | 0 | 2 | 0

46. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 29
Description: as for outcome 28
Time Frame: At Day 29 (28 days after the first study intervention administration) compared to Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 45 | 15
Participants
  ALT: Below (baseline) - below (Day 29) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 29) | 3 | 1 | 0
  ALT: Above (baseline) - below (Day 29) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 29) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 29) | 35 | 31 | 12
  ALT: Above (baseline) - within (Day 29) | 5 | 5 | 2
  ALT: Below (baseline) - above (Day 29) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 29) | 2 | 6 | 1
  ALT: Above (baseline) - above (Day 29) | 0 | 2 | 0
  AST: Below (baseline) - below (Day 29) | 1 | 0 | 0
  AST: Within (baseline) - below (Day 29) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 29) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 29) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 29) | 39 | 41 | 11
  AST: Above (baseline) - within (Day 29) | 3 | 0 | 1
  AST: Below (baseline) - above (Day 29) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 29) | 1 | 2 | 1
  AST: Above (baseline) - above (Day 29) | 1 | 2 | 2
  Creatinine: Below (baseline) - below (Day 29) | 3 | 2 | 1
  Creatinine: Within (baseline) - below (Day 29) | 1 | 0 | 0
  Creatinine: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 29) | 0 | 1 | 0
  Creatinine: Within (baseline) - within (Day 29) | 41 | 42 | 14
  Creatinine: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 29) | 4 | 3 | 3
  Blood Urea Nitrogen: Within (baseline) - below (Day 29) | 8 | 6 | 3
  Blood Urea Nitrogen: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 29) | 8 | 9 | 1
  Blood Urea Nitrogen: Within (baseline) - within (Day 29) | 25 | 27 | 8
  Blood Urea Nitrogen: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 29) | 45 | 44 | 15
  Basophils: Above (baseline) - within (Day 29) | 0 | 1 | 0
  Basophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 29) | 45 | 45 | 15
  Eosinophils: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 29) | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 29) | 1 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 29) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 29) | 38 | 39 | 12
  Hemoglobin: Above (baseline) - within (Day 29) | 0 | 1 | 0
  Hemoglobin: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 29) | 1 | 2 | 1
  Hemoglobin: Above (baseline) - above (Day 29) | 4 | 3 | 2
  Lymphocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 29) | 44 | 44 | 13
  Lymphocytes: Above (baseline) - within (Day 29) | 1 | 0 | 2
  Lymphocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 29) | 0 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 29) | 44 | 45 | 15
  Monocytes: Above (baseline) - within (Day 29) | 0 | 0 | 0
  Monocytes: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 29) | 1 | 0 | 0
  Monocytes: Above (baseline) - above (Day 29) | 0 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 29) | 1 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 29) | 41 | 43 | 15
  Neutrophils: Above (baseline) - within (Day 29) | 1 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 29) | 2 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 29) | 0 | 1 | 0
  Platelets: Below (baseline) - below (Day 29) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 29) | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 29) | 0 | 0 | 0
  Platelets: Below (baseline) - within (Day 29) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 29) | 39 | 36 | 12
  Platelets: Above (baseline) - within (Day 29) | 2 | 2 | 0
  Platelets: Below (baseline) - above (Day 29) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 29) | 1 | 1 | 0
  Platelets: Above (baseline) - above (Day 29) | 2 | 5 | 3
  White Blood Cells [WBC]: Below (baseline) - below (Day 29) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 29) | 0 | 0 | 1
  White Blood Cells [WBC]: Above (baseline) - below (Day 29) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 29) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 29) | 43 | 43 | 13
  White Blood Cells [WBC]: Above (baseline) - within (Day 29) | 0 | 2 | 1
  White Blood Cells [WBC]: Below (baseline) - above (Day 29) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 29) | 1 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 29) | 1 | 0 | 0

47. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 85
Description: as for outcome 29
Time Frame: At Day 85 (28 days after the second study intervention administration) compared to Baseline (Day 57)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 45 | 43 | 15
Participants
  ALT: Below (baseline) - below (Day 85) | 1 | 0 | 0
  ALT: Within (baseline) - below (Day 85) | 0 | 1 | 0
  ALT: Above (baseline) - below (Day 85) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 85) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 85) | 39 | 33 | 13
  ALT: Above (baseline) - within (Day 85) | 2 | 6 | 2
  ALT: Below (baseline) - above (Day 85) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 85) | 2 | 3 | 0
  ALT: Above (baseline) - above (Day 85) | 1 | 0 | 0
  AST: Below (baseline) - below (Day 85) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 85) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 85) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 85) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 85) | 40 | 36 | 12
  AST: Above (baseline) - within (Day 85) | 2 | 2 | 1
  AST: Below (baseline) - above (Day 85) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 85) | 1 | 3 | 0
  AST: Above (baseline) - above (Day 85) | 2 | 2 | 2
  Creatinine: Below (baseline) - below (Day 85) | 3 | 4 | 1
  Creatinine: Within (baseline) - below (Day 85) | 3 | 1 | 1
  Creatinine: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 85) | 0 | 3 | 0
  Creatinine: Within (baseline) - within (Day 85) | 39 | 35 | 13
  Creatinine: Above (baseline) - within (Day 85) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 85) | 0 | 0 | 0
  Creatinine: Above (baseline) - above (Day 85) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 85) | 9 | 4 | 3
  Blood Urea Nitrogen: Within (baseline) - below (Day 85) | 3 | 6 | 1
  Blood Urea Nitrogen: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 85) | 6 | 3 | 3
  Blood Urea Nitrogen: Within (baseline) - within (Day 85) | 27 | 30 | 8
  Blood Urea Nitrogen: Above (baseline) - within (Day 85) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 85) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 85) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 85) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 85) | 43 | 43 | 15
  Basophils: Above (baseline) - within (Day 85) | 1 | 0 | 0
  Basophils: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 85) | 1 | 0 | 0
  Basophils: Above (baseline) - above (Day 85) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 85) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 85) | 41 | 43 | 15
  Eosinophils: Above (baseline) - within (Day 85) | 1 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 85) | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 85) | 3 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 85) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 85) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 85) | 36 | 38 | 12
  Hemoglobin: Above (baseline) - within (Day 85) | 1 | 2 | 0
  Hemoglobin: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 85) | 2 | 0 | 1
  Hemoglobin: Above (baseline) - above (Day 85) | 4 | 3 | 2
  Lymphocytes: Below (baseline) - below (Day 85) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 85) | 43 | 42 | 15
  Lymphocytes: Above (baseline) - within (Day 85) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 85) | 2 | 1 | 0
  Lymphocytes: Above (baseline) - above (Day 85) | 0 | 0 | 0
  Monocytes: Below (baseline) - below (Day 85) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 85) | 44 | 42 | 15
  Monocytes: Above (baseline) - within (Day 85) | 1 | 0 | 0
  Monocytes: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 85) | 0 | 0 | 0
  Monocytes: Above (baseline) - above (Day 85) | 0 | 1 | 0
  Neutrophils: Below (baseline) - below (Day 85) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 85) | 0 | 0 | 0
  Neutrophils: Above (baseline) - below (Day 85) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 85) | 41 | 41 | 14
  Neutrophils: Above (baseline) - within (Day 85) | 3 | 1 | 1
  Neutrophils: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 85) | 1 | 0 | 0
  Neutrophils: Above (baseline) - above (Day 85) | 0 | 1 | 0
  Platelets: Below (baseline) - below (Day 85) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 85) | 1 | 0 | 0
  Platelets: Above (baseline) - below (Day 85) | 1 | 0 | 0
  Platelets: Below (baseline) - within (Day 85) | 0 | 0 | 0
  Platelets: Within (baseline) - within (Day 85) | 33 | 37 | 12
  Platelets: Above (baseline) - within (Day 85) | 3 | 1 | 1
  Platelets: Below (baseline) - above (Day 85) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 85) | 3 | 1 | 0
  Platelets: Above (baseline) - above (Day 85) | 3 | 4 | 2
  White Blood Cells [WBC]: Below (baseline) - below (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 85) | 42 | 43 | 15
  White Blood Cells [WBC]: Above (baseline) - within (Day 85) | 3 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 85) | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 85) | 0 | 0 | 0

48. Primary Outcome: Stage 2: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 197
Description: as for outcome 30
Time Frame: At Day 197 (28 days after the third study intervention administration) compared to Baseline (Day 169)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
Number analyzed (Participants) | 42 | 38 | 14
Participants
  ALT: Below (baseline) - below (Day 197) | 0 | 0 | 0
  ALT: Within (baseline) - below (Day 197) | 0 | 0 | 0
  ALT: Above (baseline) - below (Day 197) | 0 | 0 | 0
  ALT: Below (baseline) - within (Day 197) | 0 | 0 | 0
  ALT: Within (baseline) - within (Day 197) | 38 | 30 | 13
  ALT: Above (baseline) - within (Day 197) | 3 | 2 | 0
  ALT: Below (baseline) - above (Day 197) | 0 | 0 | 0
  ALT: Within (baseline) - above (Day 197) | 0 | 6 | 1
  ALT: Above (baseline) - above (Day 197) | 1 | 0 | 0
  AST: Below (baseline) - below (Day 197) | 0 | 0 | 0
  AST: Within (baseline) - below (Day 197) | 0 | 0 | 0
  AST: Above (baseline) - below (Day 197) | 0 | 0 | 0
  AST: Below (baseline) - within (Day 197) | 0 | 0 | 0
  AST: Within (baseline) - within (Day 197) | 36 | 32 | 12
  AST: Above (baseline) - within (Day 197) | 2 | 2 | 0
  AST: Below (baseline) - above (Day 197) | 0 | 0 | 0
  AST: Within (baseline) - above (Day 197) | 1 | 2 | 1
  AST: Above (baseline) - above (Day 197) | 3 | 2 | 1
  Creatinine: Below (baseline) - below (Day 197) | 4 | 4 | 1
  Creatinine: Within (baseline) - below (Day 197) | 2 | 1 | 0
  Creatinine: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Creatinine: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Creatinine: Within (baseline) - within (Day 197) | 35 | 33 | 13
  Creatinine: Above (baseline) - within (Day 197) | 0 | 0 | 0
  Creatinine: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Creatinine: Within (baseline) - above (Day 197) | 1 | 0 | 0
  Creatinine: Above (baseline) - above (Day 197) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - below (Day 197) | 4 | 3 | 3
  Blood Urea Nitrogen: Within (baseline) - below (Day 197) | 9 | 5 | 1
  Blood Urea Nitrogen: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - within (Day 197) | 8 | 2 | 1
  Blood Urea Nitrogen: Within (baseline) - within (Day 197) | 21 | 28 | 9
  Blood Urea Nitrogen: Above (baseline) - within (Day 197) | 0 | 0 | 0
  Blood Urea Nitrogen: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Blood Urea Nitrogen: Within (baseline) - above (Day 197) | 0 | 0 | 0
  Blood Urea Nitrogen: Above (baseline) - above (Day 197) | 0 | 0 | 0
  Basophils: Below (baseline) - below (Day 197) | 0 | 0 | 0
  Basophils: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Basophils: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Basophils: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Basophils: Within (baseline) - within (Day 197) | 42 | 38 | 14
  Basophils: Above (baseline) - within (Day 197) | 0 | 0 | 0
  Basophils: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Basophils: Within (baseline) - above (Day 197) | 0 | 0 | 0
  Basophils: Above (baseline) - above (Day 197) | 0 | 0 | 0
  Eosinophils: Below (baseline) - below (Day 197) | 0 | 0 | 0
  Eosinophils: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Eosinophils: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Eosinophils: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Eosinophils: Within (baseline) - within (Day 197) | 42 | 38 | 14
  Eosinophils: Above (baseline) - within (Day 197) | 0 | 0 | 0
  Eosinophils: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Eosinophils: Within (baseline) - above (Day 197) | 0 | 0 | 0
  Eosinophils: Above (baseline) - above (Day 197) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - below (Day 197) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Hemoglobin: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Hemoglobin: Below (baseline) - within (Day 197) | 1 | 0 | 0
  Hemoglobin: Within (baseline) - within (Day 197) | 28 | 29 | 6
  Hemoglobin: Above (baseline) - within (Day 197) | 6 | 2 | 3
  Hemoglobin: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Hemoglobin: Within (baseline) - above (Day 197) | 1 | 1 | 1
  Hemoglobin: Above (baseline) - above (Day 197) | 5 | 6 | 4
  Lymphocytes: Below (baseline) - below (Day 197) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Lymphocytes: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Lymphocytes: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - within (Day 197) | 39 | 37 | 14
  Lymphocytes: Above (baseline) - within (Day 197) | 1 | 1 | 0
  Lymphocytes: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Lymphocytes: Within (baseline) - above (Day 197) | 1 | 0 | 0
  Lymphocytes: Above (baseline) - above (Day 197) | 1 | 0 | 0
  Monocytes: Below (baseline) - below (Day 197) | 0 | 0 | 0
  Monocytes: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Monocytes: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Monocytes: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Monocytes: Within (baseline) - within (Day 197) | 39 | 37 | 14
  Monocytes: Above (baseline) - within (Day 197) | 1 | 1 | 0
  Monocytes: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Monocytes: Within (baseline) - above (Day 197) | 1 | 0 | 0
  Monocytes: Above (baseline) - above (Day 197) | 1 | 0 | 0
  Neutrophils: Below (baseline) - below (Day 197) | 0 | 0 | 0
  Neutrophils: Within (baseline) - below (Day 197) | 0 | 1 | 0
  Neutrophils: Above (baseline) - below (Day 197) | 0 | 0 | 0
  Neutrophils: Below (baseline) - within (Day 197) | 0 | 0 | 0
  Neutrophils: Within (baseline) - within (Day 197) | 42 | 33 | 14
  Neutrophils: Above (baseline) - within (Day 197) | 0 | 1 | 0
  Neutrophils: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Neutrophils: Within (baseline) - above (Day 197) | 0 | 2 | 0
  Neutrophils: Above (baseline) - above (Day 197) | 0 | 1 | 0
  Platelets: Below (baseline) - below (Day 197) | 1 | 0 | 0
  Platelets: Within (baseline) - below (Day 197) | 0 | 0 | 0
  Platelets: Above (baseline) - below (Day 197) | 1 | 0 | 0
  Platelets: Below (baseline) - within (Day 197) | 0 | 1 | 0
  Platelets: Within (baseline) - within (Day 197) | 33 | 28 | 11
  Platelets: Above (baseline) - within (Day 197) | 4 | 5 | 0
  Platelets: Below (baseline) - above (Day 197) | 0 | 0 | 0
  Platelets: Within (baseline) - above (Day 197) | 2 | 0 | 1
  Platelets: Above (baseline) - above (Day 197) | 1 | 4 | 2
  White Blood Cells [WBC]: Below (baseline) - below (Day 197) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - below (Day 197) | 0 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - below (Day 197) | 0 | 0 | 0
  White Blood Cells [WBC]: Below (baseline) - within (Day 197) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - within (Day 197) | 41 | 36 | 14
  White Blood Cells [WBC]: Above (baseline) - within (Day 197) | 0 | 1 | 0
  White Blood Cells [WBC]: Below (baseline) - above (Day 197) | 0 | 0 | 0
  White Blood Cells [WBC]: Within (baseline) - above (Day 197) | 1 | 0 | 0
  White Blood Cells [WBC]: Above (baseline) - above (Day 197) | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAEs and All-cause mortality were reported from Day 1 to Day 337 (end of study), solicited AEs were reported from Day 1 to Day 7, Day 57 to Day 63 and Day 169 to Day 175, and unsolicited AEs were reported from Day 1 to Day 28, Day 57 to Day 84 and Day 169 to Day 196. Laboratory abnormalities were reported as change from baseline to 7 days post-vaccination (Day 8, Day 64 and Day 176 respectively) and 28 days post-vaccination (Day 29, Day 85 and Day 197 respectively).
Description: SAEs, solicited AEs and unsolicited AEs were reported for the Exposed set.
Arm/Group | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group | Stage 1: iNTS-TCV Full Dose Group | Stage 1: iNTS-GMMA + TCV Full Dose Group | Stage 1: Placebo Group | Stage 2: iNTS-TCV Full Dose Group | Stage 2: iNTS-GMMA + TCV Full Dose Group | Stage 2: Control Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/16 | 0/16 | 0/10 | 0/45 | 0/45 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/16 | 1/16 | 0/10 | 0/45 | 2/45 | 1/15
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 16/16 | 16/16 | 9/10 | 43/45 | 45/45 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group (N=4) | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group (N=4) | Stage 1: iNTS-TCV Full Dose Group (N=16) | Stage 1: iNTS-GMMA + TCV Full Dose Group (N=16) | Stage 1: Placebo Group (N=10) | Stage 2: iNTS-TCV Full Dose Group (N=45) | Stage 2: iNTS-GMMA + TCV Full Dose Group (N=45) | Stage 2: Control Group (N=15)
Malaria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: Invasive Nontyphoidal Salmonella (iNTS)-Typhoid Conjugate Vaccine (TCV) Low Dose Group (N=4) | Stage 1: iNTS-Generalized Modules for Membrane Antigens (GMMA) + TCV Low Dose Group (N=4) | Stage 1: iNTS-TCV Full Dose Group (N=16) | Stage 1: iNTS-GMMA + TCV Full Dose Group (N=16) | Stage 1: Placebo Group (N=10) | Stage 2: iNTS-TCV Full Dose Group (N=45) | Stage 2: iNTS-GMMA + TCV Full Dose Group (N=45) | Stage 2: Control Group (N=15)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 1 (1) | 0 (0) | 8 (13) | 7 (12) | 0 (0) | 6 (7) | 10 (19) | 1 (1)
Administration site pain (General disorders) | 4 (15) | 4 (13) | 16 (44) | 16 (54) | 8 (19) | 40 (145) | 45 (180) | 13 (39)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 1 (1) | 1 (1) | 6 (8) | 3 (5) | 0 (0) | 13 (23) | 15 (40) | 2 (4)
Administration site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 4 (5) | 10 (18) | 12 (24) | 3 (3) | 31 (59) | 30 (62) | 6 (10)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site hyperaesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 13 (17) | 15 (20) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 8 (9) | 8 (8) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (5) | 4 (7) | 0 (0) | 21 (36) | 20 (37) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (3) | 9 (15) | 11 (20) | 1 (1) | 29 (58) | 31 (60) | 6 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (4) | 8 (15) | 11 (19) | 4 (4) | 38 (70) | 35 (77) | 8 (12)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 3 (5) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Vaccination site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 7 (7) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT05480800/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT05480800/SAP_001.pdf